# Status Page

# PROTOCOL 14-056

# **Closed to New Accrual**

Closure Effective Date: 03/30/2016 No new subjects may be enrolled in the study as described above. Any questions regarding this closure should be directed to the study's Principal Investigator Date Submitted: [12/22/14]
Date Posted: [01/08/15]

# Alert Page

DF/HCC Protocol #: 14-056

Protocol Clarifications (non-drug related e.g. eligibility criteria, study assessments)

# **Protocol Section 9, Study Calendars:**

# Monitoring phase:

- Patient Global Impressions- Fatigue (PGI-F) should be completed at baseline visit. This will be clarified in a future protocol amendment.
- PHQ-9 and FACT-B/ES should be completed at week 4 and week 8. This
  will be clarified in a future protocol amendment.
- (+/-) 7 day window applies to all weekly monitoring visits. This will be clarified in a future protocol amendment.

# Intervention phase:

- Patient Global Impressions- Improvement (PGI-I) should be completed in place of PGI-F at week 0 randomization visit and week 5 Rx visit. This will be clarified in a future protocol amendment.
- (+/-) 7 day window applies to all visits. This will be clarified in a future protocol amendment.

Revised: 07.01.13

Local Protocol #: 14-056

# TITLE: Phase II Double-Blind Randomized Controlled Trial of Naltrexone for Treatment-Emergent Fatigue in Patients Receiving Radiation Therapy for Breast Cancer

**Coordinating Center:** Dana-Farber Cancer Institute

\*Principal Investigator (PI): Fremonta Meyer, MD

Psychosocial Oncology and Palliative Care

Dana-Farber Cancer Institute/Brigham and Women's Hospital

flmeyer@partners.org

**Other Investigators:** Alphonse Taghian, MD PhD (MGH site PI)

Radiation Oncology

Massachusetts General Hospital

ataghian@partners.org

David Fisher, MD PhD (PI of Grant)

Dermatology

Massachusetts General Hospital

dfisher3@partners.org

Hadine Joffe, MD, MSc

Psychosocial Oncology and Palliative Care

Dana-Farber Cancer Institute

hjoffe@partners.org

Kelly Irwin, MD

Psychiatry (Psycho-oncology) Massachusetts General Hospital

keirwin@partners.org

Ilana Braun, MD

Psychosocial Oncology and Palliative Care

Dana-Farber Cancer Institute ilana braun@dfci.harvard.edu

April Hirschberg, MD

Psychiatry (Psycho-oncology) Massachusetts General Hospital

ahirschberg@partners.org

Julia Wong, MD Radiation Oncology

Dana-Farber Cancer Institute

jwong@lroc.harvard.edu

# Statistician:

Andrzej Niemierko Radiation Oncology Massachusetts General Hospital aniemierko@partners.org

NCI-Supplied Agent(s): Not applicable Other Agent(s): Naltrexone or Placebo

**IND** #: IND exempt

IND Sponsor: Fremonta Meyer, MD / FDA

Protocol Version # / Version Date: Version 12 / May 3, 2018

# **SCHEMA**

# Protocol Schema





# **TABLE OF CONTENTS**

| SCE | IEMA | | iii |
|---|---|---|---|
| 1. | OBJ | ECTIVES | 1 |
| | 1.1 | Study Design | |
| | 1.2 | Primary Objectives | |
| | 1.3 | Secondary Objectives | |
| 2. | BAC | KGROUND | 3 |
| | 2.1 | Study Disease(s) | |
| | 2.2 | Drug Information | |
| | 2.3 | Rationale | |
| | 2.4 | Correlative Studies Background | 6 |
| 3. | PAR | TICIPANT SELECTION | 7 |
| | 3.1 | Eligibility Criteria for Monitoring Phase | 7 |
| | 3.2 | Exclusion Criteria for Monitoring Phase | 7 |
| | 3.3 | Eligibility Criteria for Randomization Phase | |
| | 3.4 | Exclusion Criteria | 8 |
| | 3.5 | Inclusion of Women and Minorities | 8 |
| 4. | Recruitment and REGISTRATION PROCEDURES | | |
| | 4.1 | Patient Recruitment | |
| | 4.2 | General Guidelines for DF/HCC and DF/PCC Institutions | |
| | 4.3 | Registration Process for DF/HCC and DF/PCC Institutions | 9 |
| 5. | TRE | ATMENT PLAN | 10 |
| | 5.1 | Treatment Regimen | 10 |
| | 5.2 | Pre-Treatment Criteria | 11 |
| | 5.3 | Agent Administration | 11 |
| | 5.4 | General Concomitant Medication and Supportive Care Guidelines | 12 |
| | 5.5 | Duration of Therapy | 13 |
| | 5.6 | Duration of Follow Up | 13 |
| | 5.7 | Criteria for Removal from Study | 13 |
| | 5.8 | DOSING DELAYS/DOSE MODIFICATIONS | 15 |
| 6. | ADVERSE EVENTS: LIST AND REPORTING REQUIREMENTS | | |
| | 6.1 | Expected Toxicities | 16 |
| | 6.2 | Adverse Event Characteristics | 18 |
| | 6.3 | Expedited Adverse Event Reporting | |
| | 6.4 | Expedited Reporting to Hospital Risk Management | |
| | 6.5 | Routine Adverse Event Reporting | 19 |
| 7. | PHA | RMACEUTICAL INFORMATION | |
| | 7 1 | Naltreyone | 20 |

| 8. | BIOMARKER, CORRELATIVE, AND SPECIAL STUDIES21 | |
|-----|-----------------------------------------------|--------------|
| 9. | STUDY CALENDARS | 22 |
| 10. | MEASUREMENT OF EFFECT | 26 |
| | 10.1 Other Response Parameters | 26 |
| 11. | DATA REPORTING / REGULATORY REQ | OUIREMENTS28 |
| | | 28 |
| | 11.2 Data Safety Monitoring | 28 |
| | 11.3 Multicenter Guidelines | 28 |
| | | 29 |
| 12. | STATISTICAL CONSIDERATIONS | 29 |
| | | 29 |
| | | 29 |
| | 12.3 Stratification Factors | 30 |
| | | 30 |
| | 12.5 Reporting and Exclusions | 30 |
| 13. | PUBLICATION PLAN | 31 |

#### 1. OBJECTIVES

The objective of this study is to determine whether the opioid antagonist naltrexone reduces radiation therapy-related fatigue more than placebo does in patients undergoing radiotherapy for breast cancer.

## 1.1 Study Design

A randomized, double-blind, parallel-arm 5-week clinical trial will be used to determine the effect of naltrexone on fatigue emerging during radiation therapy for non-metastatic breast cancer (see Protocol Schema). The trial has two phases (a monitoring phase and an intervention phase) requiring two separate consents.

Monitoring phase: Prior to initiating radiotherapy, participants will be approached and consented for the monitoring phase of the study, which involves longitudinal monitoring of fatigue in order to establish whether a patient develops fatigue after starting radiation. The level of preradiotherapy fatigue will be obtained during the final 3 weeks before, or within 3 days, that radiotherapy is started. Participants who provide baseline data and report suicidal ideation either spontaneously or on a self-report questionnaire will be excluded from subsequent weekly monitoring of fatigue. All other participants will undergo weekly monitoring of fatigue via a brief self-report questionnaire (Functional Assessment of Chronic Illness Therapy-Fatigue Subscale; FACIT-F) once radiation therapy begins. Those whose fatigue symptoms increase above the pre-specified threshold at any point during the monitoring period will be approached about enrollment into the intervention phase of the study. The monitoring period will continue up until one month after the conclusion of radiotherapy. Radiation oncologists will refer potentially eligible patients to the monitoring phase of the study. The clinical research coordinator will be trained to administer the screening consent and will follow participants during the monitoring phase of the study and notify the radiation oncologist if fatigue emerges/worsens after radiation therapy has begun, so that participation in the intervention phase of the study can be discussed with these patients.

Intervention phase: Radiation oncologists will consent patients who develop treatment-emergent fatigue developing during or within one month after completion of radiation therapy and who are interested in participating in the intervention phase of the study. After informed consent is obtained and final eligibility determination is complete, participants will have 5 study visits: one at study entry to initiate treatment (week 0), one to rule out any contraindication to the scheduled dose escalation (week 1), one at the conclusion of medication treatment for treatment outcome assessment and safety monitoring (week 5), and the last at four weeks after discontinuation of study drug vs. placebo (week 9). All intervention visits have a window of  $\pm$  7 days.

<u>Study treatment</u>: The treatment schedule includes a daily dose of double-blinded naltrexone vs. placebo for 5 weeks. Treatment will be initiated at 25 mg/day (or equivalent placebo) during the first week to improve tolerability. The dose will be escalated to 50 mg/day (or equivalent placebo) after one week barring significant early improvement in fatigue or adverse events precluding dose escalation, and participants will continue to take 50 mg/day (or 25 mg/day if dose is not escalated) for 4 weeks to complete a 5-week treatment period.



# 1.2 Primary Objectives

To determine the effect of naltrexone on treatment-emergent fatigue during radiation therapy for breast cancer. The primary comparison is between changes in fatigue scores in the naltrexoneversus the placebo-treated participants as measured by the FACIT-F subscale.

# 1.3 Secondary Objectives

- 1.3.1. To determine the effect of naltrexone on exploratory outcomes including: mood, anxiety, subjective cognitive function, sleep, pain, and quality of life, and the extent to which changes in fatigue correlate with changes in these symptom endpoints. These outcomes have been shown to be associated with cancer fatigue in prior studies involving breast cancer patients<sup>1</sup> <sup>2-4</sup>.
- 1.3.2. To determine the course, predictors, and correlates of fatigue during radiotherapy for breast cancer in a large controlled sample

### 2. BACKGROUND

## 2.1 Study Disease(s)

Fatigue is one of the most common side effects of both radiation therapy and chemotherapy. It is the greatest predictor of poor quality of life in cancer patients undergoing treatment, and very often results in an inability to perform activities of daily living easily accomplished prior to treatment (Hickok et al., 1996). More importantly, severe fatigue can result in breaks in treatment that adversely affect treatment efficacy and ultimately compromise survival.

Despite its importance as a side effect that impairs quality of life and reduces treatment adherence, treatment options for cancer-related fatigue are limited. Exercise programs and psychological interventions such as cognitive-behavioral therapy appear to have a positive effect on cancer-related fatigue<sup>5</sup>, but are not accessible or feasible for all patients who might benefit. In terms of pharmacologic strategies, a recent meta-analytic review suggested that stimulants (e.g., methylphenidate) and hematopoietic agents (the latter only in the presence of anemia) may be effective<sup>6</sup>. However, the effect size of stimulants, albeit clinically significant, is small; hematopoietic agents such as erythropoietin are less widely used given associated increase in risk for thrombovascular events and mortality. Modafinil and armodafinil, both non-amphetamine based stimulant-like medications that improve fatigue related to obstructive sleep apnea and multiple sclerosis, have been the focus of more recent randomized trials. Specifically, a Phase III trial in patients with a wide variety of cancer types found that modafinil has significantly positive effects for severe, but not mild to moderate, cancer fatigue<sup>7</sup>. Trial durations for effective pharmacological interventions in cancer fatigue are variable, ranging from 2-12 weeks, many of which show benefit with 4 weeks.<sup>6</sup>

Although their use is widespread, stimulants and stimulant-like medications may exert nonspecific effects that are not tied to an underlying cancer-related mechanism of fatigue. Some work has suggested that cancer fatigue may be driven by the activation of pro-inflammatory cytokines, paving the way for study of cytokine inhibitors such as eternacept, which in a study of advanced cancer patients on chemotherapy appeared to reduce fatigue<sup>8</sup>. Other proposed mechanisms include disruptions in the hypothalamic-pituitary-adrenal axis, as shown by studies revealing altered cortisol responses in fatigued cancer survivors<sup>9</sup> and metastatic breast cancer patients<sup>10</sup>. However, at this point, there is limited direct clinical evidence to substantiate these theories. Thus, interventions to manage cancer-related fatigue continue to be empirical in nature, possibly accounting for their modest effect sizes.

The present study stems from a preclinical observation implicating upregulation of the endogenous opioid system as a potential underlying mechanism for fatigue in patients receiving radiotherapy. As in humans, irradiation (of the tail) has been shown to induce lethargy in rodent models and beta-endorphin levels increase in response to tail irradiation. Dr. Fisher's lab has observed that the opiate receptor antagonist naloxone reverses fatigue induced by irradiation. Preclinical data (further described in Section 2.3, Rationale) suggest that the elevations in beta-endorphin may be responsible for radiation-related fatigue, and that pharmacologic treatment with a mu-opioid receptor antagonist may ameliorate the fatigue symptoms. Thus, the primary aim of this study is to determine whether the widely used and FDA-approved opioid antagonist naltrexone might reduce radiation-emergent fatigue in humans.

Given results of pre-clinical studies, naltrexone is a viable treatment to investigate for

radiation-related fatigue in cancer patient populations who are not expected to require opioid therapy. Breast cancer patients receiving radiotherapy represent an important population to study because fatigue develops commonly during radiotherapy and concurrent therapy with opioids is rare. Notably, existing literature provides widely variable estimates (38-75%) of the prevalence of breast radiotherapy-emergent fatigue<sup>11,12</sup> as well as differing evidence as to the most important predictors of fatigue in this population. Longitudinal studies have found that fatigue levels gradually increase during a course of breast radiotherapy, particularly during the first four weeks of treatment. 13-15 Several studies have investigated clinical correlates of radiation-related fatigue in this population. Donovan found that patients (N=134) pre-treated with chemotherapy reported less fatigue during radiotherapy as compared to patients who did not receive chemotherapy, and that demographic and disease-related variables did not predict the extent of fatigue; however, psychological variables were not examined in this study. <sup>16</sup> Manir described anemia as the most important predictor of fatigue (N=72)<sup>12</sup> whereas other studies have found no relationship between hemoglobin levels and fatigue.<sup>13</sup> Recently, Taunk compared different radiotherapeutic regimens for early-stage breast cancer (overall N=80) and suggested that partial breast irradiation may reduce fatigue as compared to hypofractionated and standard whole breast irradiation.<sup>17</sup> However, in the largest cohort study to date (N=250), Reidunsdatter identified medical comorbidity as a more important determinant of increased fatigue during breast radiotherapy than radiotherapy type. 18 By contrast, Courtier reported that anxiety, elevated pre-treatment fatigue, and diagnoses other than invasive ductal carcinoma (e.g. DCIS or lobular subtypes) predicted radiation-emergent fatigue (N=100). 11 More study of the clinical correlates and course of fatigue during radiotherapy is warranted in the breast cancer population given the relatively small sample sizes, variable inclusion of relevant medical and psychosocial variables in models to predict fatigue, and conflicting findings to date. The monitoring phase of the present study offers an embedded opportunity to analyze the course, predictors, and correlates of radiotherapyrelated fatigue in a controlled breast cancer population.

# 2.2 Drug Information

### Mechanism of Action

Naltrexone hydrochloride is a competitive antagonist at mu and delta opioid receptors. As such, it blocks the binding of beta-endorphin to the mu opioid receptor. Although naltrexone has been shown to have variable effects on beta-endorphin levels<sup>19-21</sup>, endorphin levels do not predict opioid activity in the presence of a mu opioid receptor antagonist like naltrexone.

## Clinical Studies

In human studies, naltrexone has been effective in decreasing both use and cravings in patients with alcohol and opioid dependence<sup>22,23</sup> Naltrexone (in both oral and long-acting injectable IM formulations) is currently FDA approved for the treatment of alcohol and opioid dependence. Off-label studies have shown efficacy of naltrexone (in combination with bupropion) in causing significant weight loss in patients with uncomplicated obesity<sup>24</sup>. The agent has also been studied off-label for treatment of binge eating disorder and self-injurious behavior. The placebo-controlled studies that demonstrated the efficacy of naltrexone as an adjunctive treatment of alcoholism (in patients > 18 years of age) used a dose regimen of 50 mg po daily for up to 12 weeks; doses effective for obesity were somewhat lower (16-32mg). Clinically, the standard, widely-utilized, dose, attained in the vast majority of patients with alcohol and opioid

dependence, is 50mg daily. Furthermore, prior research suggests that women achieve higher serum levels of naltrexone than men, and that women are significantly less adherent to 100mg doses (due to decreased tolerability) than to placebo or 25-50mg doses <sup>25</sup>.

The durations of most placebo-controlled trials of naltrexone for alcohol and opioid dependence have ranged from 12-52 weeks, although shorter positive trials (3-12 weeks) exist in the literature. Clinically, for treatment of alcohol and opioid dependence, an initial 4-month course of naltrexone is recommended, and the medication can be continued indefinitely in the setting of good response. The present study differs in that the target population will receive naltrexone for radiotherapy-emergent fatigue, which has been shown in prior studies to improve spontaneously after the conclusion of radiation treatment, returning to pre-treatment levels in the majority of patients by three months after radiotherapy. Therefore, a 5-week trial duration will be utilized in order to minimize the possibility of missing the appropriate time period in which to demonstrate treatment effect as opposed to spontaneous recovery. Further supporting the 5-week trial duration is the observation that patients often demonstrate therapeutic benefit from naltrexone within the first few days or weeks of treatment.

### **Pharmacokinetics**

Naltrexone has a volume of distribution of 1350 L, and is 21% protein bound. It is metabolized hepatically via dihydrodiol dehydrogenase and conjugation to its principal metabolite, 6-beta-naltrexol. It is 53-75% renally excreted, mostly as metabolites, less than 2% unchanged. The elimination half-life of 6-beta-naltrexone is 5-10 days.

Despite its hepatic metabolism, naltrexone does not interact with the cytochrome P450 enzyme system.

### 2.3 Rationale

## Radiation Therapy

The majority of cancer patients receiving radiation therapy are treated with fractionated external beam radiation, in which a daily dose of radiation from an external source targets a tumor within the body. A significant portion of patients receiving external beam radiation experience fatigue three to four weeks into a typical five- to eight-week radiation course, regardless of the location of the tumor or the radiation field. This fatigue usually lasts for approximately three weeks after treatment and either resolves spontaneously, or can persist for weeks to months.

Interestingly, patients receiving radiation that targets only superficial structures (i.e. breast cancer patients) can become equally as fatigued as patients receiving radiation to deeper structures, and fatigue is more highly correlated with skin dose and field size than with depth of radiation<sup>28,29</sup>. In fact, the one commonality among radiation therapy regimens that cause fatigue is that there is a significant skin dose. This led us to hypothesize that factors produced in the skin in response to radiation may play a role in radiation-induced fatigue.

DNA damage resulting from radiation exposure causes upregulation of expression of p53 dependent genes in skin cells. One recently-identified p53-dependent gene upregulated in keratinocytes in response to radiation exposure encodes a long-lived endogenous opioid called  $\beta$ -

endorphin<sup>30</sup>. B-endorphin induction following radiation exposure was observed during studies elucidating the pathway through which ultraviolet radiation stimulates skin pigmentation (tanning). In the pigmentation response following ultraviolet radiation exposure, there is a p53induced expression of pro-opiomelanocortin (POMC) in keratinocytes. POMC is cleaved into various biologically-functional peptides. One of these peptides, Melanocyte Stimulating Hormone (MSH), is important in the tanning response, acting in a paracrine fashion to stimulate melanocytes to produce pigment. Another peptide derived from POMC production and cleavage following multiple types of DNA damage is the endogenous opioid β-endorphin. Opioid drugs (such as morphine) often cause fatigue and lethargy when they are used to treat pain. Dr. Fisher's data in mice show that plasma β-endorphin levels are elevated significantly by 3 weeks into a 6week regimen of daily tail radiation that models radiation therapy in cancer patients receiving radiation to superficial structures. In contrast to humans, mice do not exhibit fatigue in response to exogenous administration of opiate drugs<sup>31</sup>. However, quantitative behavioral studies indicated significant changes in phenotypes associated with morphine administration, including mechanical and thermal nociception, in tail-irradiated mice that did not occur in non-irradiated mock-treated counterparts. Furthermore, these changes were reversed upon administration of the opioid antagonist naloxone. In these tail-irradiated mice, β-endorphin plasma levels diminish over the 4 weeks following the end of the radiation regimen.

# Chemotherapy

Patients receiving chemotherapy typically become debilitatingly fatigued, even more predictably than radiation therapy patients. As mentioned above, the increased production of  $\beta$ -endorphin following radiation exposure-induced DNA damage is a p53-dependent process. Many common chemotherapeutics are DNA damaging agents that induce p53, and therefore p53-dependent genes, to cause apoptosis of cancer cells<sup>32</sup>. As transcription of the gene encoding  $\beta$ -endorphin is responsive to p53, it is thus plausible that the fatigue caused in patients receiving chemotherapy is the result of increased  $\beta$ -endorphin production following chemotherapy-induced p53 up-regulation in target cells. A treatment that blocked the effects of  $\beta$ -endorphin might then also reduce any residual fatigue from chemotherapy.

### 2.4 Correlative Studies Background

At the blood draw obtained for eligibility determination immediately prior to randomization, whole blood samples will be banked for analysis of OPRM1 (mu opioid receptor) genetic variants, specifically the Asn40Asp missense variant which has a frequency of 0.10-0.15 in Caucasians, 0.21 in Ashkenazi Jews, 0.25-0.45 in East Asians, and 0.14 in Hispanics.<sup>33</sup> The Asn40Asp variant has been shown to bind beta-endorphin approximately three times more tightly than the most common allelic form of the receptor,<sup>34</sup> and it has predicted good clinical response to naltrexone in alcohol and opioid dependence.<sup>33,35,36</sup>

Banked specimens will also be available for future exploratory examination of proinflammatory biomarkers such as expression-regulating polymorphisms in pro-inflammatory cytokine genes, which in recent studies have correlated with increased fatigue severity, depressive symptoms and memory complaints.<sup>37</sup>

### 3. PARTICIPANT SELECTION

# 3.1 Eligibility Criteria for Monitoring Phase

- 3.1.1 Age  $\geq 18$
- 3.1.2 Diagnosis of: invasive breast cancer (stage I-III), ductal carcinoma in situ, lobular carcinoma in situ, lobular carcinoma
- 3.1.3 Plan to receive radiation therapy, or within 3 days of starting radiation therapy
- 3.2 Exclusion Criteria for Monitoring Phase
- 3.2.1 Suicidal ideation, as determined via PHQ-9
- 3.2.2 Non-English speaking

# 3.3 Eligibility Criteria for Randomization Phase

- 3.3.1 Participants may have had prior breast surgery and/or chemotherapy.
- 3.3.2 Age  $\geq$ 18 years.

Because no dosing or adverse event data are currently available on the use of naltrexone in cancer patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.

3.3.3 Participants must have acceptable pre-treatment laboratory values as defined below:

- total bilirubin within normal institutional limits

- AST(SGOT)/ALT(SGPT)  $\leq 2.5 \times \text{institutional upper limit of normal}$ 

- creatinine within normal institutional limits

 $\cap R$ 

- creatinine clearance >60 mL/min/1.73 m<sup>2</sup> for patients with creatinine levels

above institutional normal.

- TSH <10 mIU/L

- 3.3.4 If child-bearing potential, willingness to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
- 3.3.5 Ability to understand and the willingness to sign a written informed consent document

- 3.3.6 Receiving radiation therapy of any type at DFCI, BWH, MGH, or affiliated network sites (including but not limited to partial breast irradiation, two-field, three-field, and four-field plans)
- 3.3.7 FACIT-F subscale score >=10 pre-radiation therapy and decrease in FACIT-F of 10 points or more as compared to prior FACIT

### 3.4 Exclusion Criteria

- 3.4.1 Participants with major depressive disorder and/or suicidal ideation as determined by PHQ-9.
- 3.4.2 Participants who are receiving any other investigational agents that might interact with study medication or influence the measurement of study outcomes.
- 3.4.3 Participants with known metastatic disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
- 3.4.4 History of allergic reactions attributed to compounds of similar chemical or biologic composition to naltrexone.
- 3.4.5 Participants who have used opioid-containing medications (including cough/cold medications containing codeine and/or antidiarrheals containing loperamide) in the past 2 weeks, or who are expected to require opioid-containing medications within the duration of the treatment period.
- 3.4.6 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
- 3.4.7 Pregnant women are excluded from this study because naltrexone is category C agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with naltrexone, breastfeeding should be discontinued if the mother is treated with naltrexone.
- 3.2.8 Participants using other contraindicated medications (thioridazine, yohimbine)

### 3.5 Inclusion of Women and Minorities

Women of all races and ethnic groups are eligible for this trial.

#### 4. RECRUITMENT AND REGISTRATION PROCEDURES

### 4.1 Patient Recruitment

The study team will review radiation oncologist's schedules and Epic records for basic information to identify potential patients. With the radiation oncologist's permission, a trained individual will approach the patient to discuss this study. If a patient decides to participate in this study, written informed consent will be obtained.

### 4.2 General Guidelines for DF/HCC and DF/PCC Institutions

Institutions will register eligible participants with the DF/HCC Quality Assurance Office for Clinical Trials (QACT) central registration system. There will be a two-part registration: the 1<sup>st</sup> part for the monitoring phase of the study and the 2<sup>nd</sup> part for the intervention phase. The relevant part of the registration must be completed prior to the initiation of fatigue monitoring (1st part) and therapy (2<sup>nd</sup> part). Any participant not registered to the protocol before treatment begins will be considered ineligible and registration will be denied.

An investigator will confirm eligibility criteria and a member of the study team will complete the QACT protocol-specific eligibility checklist. The CRC will be consenting participants to monitoring phase only. Intervention phase consent will be done by an MD who is listed as a co-investigator.

Following registration, participants may begin protocol treatment. Issues that would cause treatment delays should be discussed with the Overall Principal Investigator (PI). If a participant does not receive protocol therapy following registration, the participant's registration on the study may be canceled. Notify the QACT Registrar of registration cancellations as soon as possible.

# 4.3 Registration Process for DF/HCC and DF/PCC Institutions

The QACT registration staff is accessible on Monday through Friday, from 8:00 AM to 5:00 PM Eastern Standard Time. In emergency situations when a participant must begin treatment during off-hours or holidays, call the QACT registration line at 617-632-3761 and follow the instructions for registering participants after hours.

The registration procedures are as follows:

- Obtain written informed consent from the participant prior to the performance of any protocol specific procedures or assessments.
- Complete the QACT protocol-specific eligibility checklist using the eligibility assessment documented in the participant's medical record and/or research chart. To be eligible for registration to the protocol, the participant must meet all inclusion and exclusion criterion as described in the protocol and reflected on the eligibility checklist.

<u>Reminder</u>: Confirm eligibility for ancillary studies at the same time as eligibility for the treatment protocol. Registration to both treatment and ancillary protocols will not be completed if eligibility requirements are not met for all studies.

- Fax the eligibility checklist(s) and all pages of the consent form(s) to the QACT at 617-632-2295. For Phase I protocols, attach participant dose level assignment confirmation from the sponsor.
- The QACT Registrar will (a) review the eligibility checklist, (b) register the participant on the protocol, and (c) randomize the participant when applicable. The randomization will be a block randomization at each site (DFCI/BWH vs MGH).
- An email confirmation of the registration and/or randomization will be sent to the Overall PI, study coordinator(s) from the Lead Site, treating investigator and registering person immediately following the registration and/or randomization.

### 5. TREATMENT PLAN

## 5.1 Treatment Regimen

Patients consented to the intervention phase will be randomized to naltrexone (25mg for 1 week, followed by 50mg for 4 weeks) or matching placebo. All participants will be instructed to take the double-blinded medications in the morning with food. The medication should be swallowed whole. If the patient misses or vomits a dose, they can be re-dosed within an 8-hour time frame.

The patient will be requested to maintain a medication diary of each dose of medication. The medication diary will be returned to clinic staff at the end of the study.

# **Study Plan: Randomization Phase**



<sup>&</sup>lt;sup>1</sup>Functional Assessment of Chronic Illness Therapy-Fatigue Subscale

### 5.2 Pre-Treatment Criteria

No evidence of hepatic or renal impairment and serum HCG negative, as described in the eligibility criteria above

# 5.3 Agent Administration

All participants will be instructed to swallow the double-blinded medications in the morning with food.

Monitoring and Intervention Phases: Visit Breakdown – Refer to study calendar in section 9.

# Monitoring Phase (duration: 1-10 weeks):

- Visit 1: Collection of baseline data.
  - a. Patient demographic information and clinical characteristics will be collected by self-administered surveys.

- b. Completion of self-reported fatigue, anxiety, depression, sleep and quality of life questionnaires.
- <u>Visits 2-10 (in person or by phone):</u> Monitoring procedures including completion of self-reported fatigue and other quality of life questionnaires

The occasional mis-timed (or missed) FACIT does not automatically constitute a protocol violation. However, in order to remain in compliance with the protocol, a minimum of 4 FACITs is needed for partial breast irradiation patients, 5 FACITs for hypofractionation patients, and 7 FACITs for standard (6 week) fractionation patients. The monitoring phase terminates either at entrance into the intervention phase of the study, or at 4 weeks after the conclusion of radiation therapy, whichever comes first.

# Intervention Phase (duration 5 weeks):

### • Visit 1a:

- a. consent for trial;
- b. review of concomitant medications;
- c. complete baseline fatigue questionnaire (unless completed within past week)—may be completed at Visit 1b;
- d. complete anxiety, depression, sleep and quality of life questionnaires (unless completed within past week)—may be completed at Visit 1b;
- e. urine HCG only in women with reproductive potential; blood draw to evaluate LFTs, Hct, BUN/Cr unless results are available within the previous month;
- f. specimens will be banked for future analysis of fatigue-related genetic polymorphisms and inflammatory biomarkers (participants can opt out of specimen banking)
- <u>Visit 1b</u>: laboratory study results reviewed to confirm eligibility; receive medication bottles and medication diary; receive patient education sheet on contraindicated medications and safety card (see Appendix A); <u>Visit 2</u> (one week after starting study drug vs. placebo): fatigue/response and adverse event assessment for dose escalation, review of concomitant medications, fatigue assessment
- <u>Visit 3 (five weeks after initiating study drug vs placebo):</u> complete follow-up fatigue, anxiety, depression, sleep and quality of life questionnaires; review of concomitant medications; return medication bottles and diaries. Blood draw for LFTs.

# 5.4 General Concomitant Medication and Supportive Care Guidelines

For nausea, the suggested approach based on clinical guidance is for the patient to take naltrexone with a tablespoon of simethicone (e.g., Gas-X® and Mylicon®) or bismuth subsalicylate (e.g., Pepto-Bismol).

Drug Interactions with Naltrexone:

The following medications are contraindicated because their effect may be blocked:

- Cough/cold medications: if medication contains an opioid (e.g. codeine)
- Antidiarrheal medications: if medication contains an opioid (e.g. loperamide)

Opioid analgesics: Contraindicated because greater amount of opiate analgesia may be required than usual which may result in deeper and more prolonged respiratory depression than if the patient were not taking naltrexone

Thioridazine: May result in lethargy and somnolence

Yohimbine: May result in anxiety and increased pulse and blood pressure

Nonsteroidal anti-inflammatory drugs (NSAIDs): At doses above that used in this study, may result in liver enzyme elevations (i.e., AST and ALT) in combination with regular use of very high doses of naltrexone (200–250 mg/day). This effect has only been observed above the recommended therapeutic dose range of naltrexone (i.e., >50–100 mg); therefore these medications are not considered to be contraindicated.

# 5.5 **Duration of Therapy**

Duration of therapy will be five weeks. In the absence of adverse event(s), treatment will continue for the entire five weeks unless one of the following criteria applies:

- Initiation of opioid-containing medications
- Intercurrent illness that prevents further administration of treatment
- Unacceptable adverse event(s)
- Participant demonstrates an inability or unwillingness to comply with the oral medication regimen and/or documentation requirements
- Participant decides to withdraw from the study
- General or specific changes in the participant's condition render the participant unacceptable for further treatment in the judgment of the treating investigator

### 5.6 Duration of Follow Up

Participants in the monitoring phase of the study will be followed for a maximum of 10 weeks, ending 4 weeks after cessation of radiotherapy or until they consent (if eligible) to participate in the intervention phase of the study. Those in the intervention phase will be followed until 4 weeks post-treatment. Participants removed from study for unacceptable adverse event(s) will be followed until the end of the study and beyond, until resolution or stabilization of the adverse event has occurred.

### 5.7 Criteria for Removal from Study

1. Initiation of opioid therapy, or newly expected need for opioid therapy while on study drug

- 2. Emergence of suicidal ideation
- 3. Moderate or severe hepatic impairment (AST and ALT > 3x ULN; Bilirubin > 1.5 ULN)
- 4. Moderate or severe renal impairment (Creatinine > 1.5x ULN)
- 5. Clinically significant respiratory or cardiac disease
- 6. Significant deviation from study protocol
- 7. Need to hold drug for more than 3 days, for any reason

Participants will be removed from the study when any of the criteria listed in Section 5.7 applies. The reason for study removal and the date the participant was removed must be documented in the case report form (CRF). Alternative care options will be discussed with the participant.

A QACT Treatment Ended/Off Study Form should be filled out when a participant completes study treatment and again when the participant comes off study. This form can be found on the QACT website or obtained from the QACT registration staff.

In the event of unusual or life-threatening complications, investigators must notify the Overall PI, Fremonta Meyer, MD, at 617-732-5700, pager ID 17231 or via email (<u>flmeyer@partners.org</u>) within 24 hours of discovery.

Psychiatric emergencies: Suicidal ideation is a rare (<=1%) adverse event associated with naltrexone use in individuals receiving IM naltrexone for alcohol and opioid dependence but it was not observed in those treated with naltrexone orally or in those receiving it for other indications (i.e., obesity, smoking cessation, binge eating disorder). Suicidal ideation will be assessed during the trial each time the PHQ-9 depression self-report questionnaire is completed. The CRC will be scoring the PHQ9 and if the score is greater than or equal to 10, the CRC will notify the participant's Radiation Oncologist as well as the study's psychiatrist so that they can discuss with the participant the options for clinical follow-up and further care. Suicidal ideation that is indicated on the PHQ-9 or spontaneously reported will constitute a serious adverse event. This evaluation will be conducted by one of the study clinicians with psychiatric expertise and/or by mental health staff in the MGH or BWH emergency rooms, if appropriate. These participants will be followed by study psychiatrists until a local mental health clinician is available for ongoing treatment. Study medication will be discontinued in any participant who develops suicidal ideation. The following established algorithm will be employed:

### Specific Algorithms for Addressing Participant Reports of Suicidal Ideation

#### Algorithm based on participant volunteering Algorithm based on response to *PHO-9*: possible suicidal ideation ITEM 13.9: Over the last 2 weeks, how often have you been bothered by .... Ask: Have you had thoughts of actually hurting .... Thoughts that you would be better off dead or of vourself? hurting yourself in some way? If participant responds .... (shaded areas) More than Several Nearly Not at all half the every day days days If participant responds .... (shaded area) 0 2 3 NO YES



Ask three screening questions about plan, probability and preventing factors:

### Plan:

1. Have you thought about how you might actually hurt yourself?

NO YES [ask HOW?]

### Probability:

2. There's a big difference between having a thought and acting on a thought. How likely do you think it is that you will act on these thoughts about hurting yourself or ending your life sometime over the next month?

Not at all likely Somewhat Very likely

### Preventing factors:

3. Is there anything that would prevent or keep you from harming yourself?

NO YES [ask WHAT?]

# Any shaded responses to the three screening questions requires one of the following to be done the same day:

- Refer participant to study psychiatrist
- Send participant to an emergency room, or
- Send participant to another mental health professional

### 5.8 DOSING DELAYS/DOSE MODIFICATIONS

Study drug will be increased to 50mg after 1 week of therapy unless fatigue has improved substantially on the lower dose or there are contraindications to this planned dose increase (including, but not limited to, adverse events grade II or higher that are thought to be related to study drug), as judged by the research nurse and study psychiatrist.

Some patients may tolerate the 25mg dose but develop toxicity after the dose is increased to 50mg. Hence, drug dose can be decreased from 50mg to 25mg in the setting of new-onset adverse events grade II or higher by CTCAE judged to be definitely or probably related to study drug.

Study drug (either at the 25mg or 50mg dose) can also be held for up to three days and then

# Shaded response requires one of the following to be done the same day:

- Refer participant to study psychiatrist
- Send participant to an emergency room, or
- Send participant to another mental health professional

restarted in setting of adverse events grade II or higher by CTCAE if these events are judged to be possible, unlikely or unrelated to study drug. If the drug must be held for more than three days, the participant will need to come off the study.

| | Remain at 25 mg dose instead of increasing to 50 mg | Dose reduction to 25 mg dose after increasing to 50 mg dose | Dose hold at either 25 mg or 50 mg dose for up to 3 days |
|---|---|---|---|
| Conditions | <ul> <li>Substantially reduced fatigue on 25 mg dose</li> <li>Adverse events grade II or higher determined by CTCAE guidelines</li> <li>Other conditions deemed significant by the research nurse and study psychiatrist</li> </ul> | <ul> <li>New onset adverse events grade II or higher by CTCAE guidelines definitely or probably related to study drug</li> <li>Other conditions deemed significant by the research nurse and study psychiatrist</li> </ul> | <ul> <li>Adverse events grade II or higher by CTCAE guidelines possibly, unlikely, or unrelated to study drug</li> <li>Other conditions deemed significant by the research nurse and study psychiatrist</li> </ul> |

### 6. ADVERSE EVENTS: LIST AND REPORTING REQUIREMENTS

Adverse event (AE) monitoring and reporting is a routine part of every clinical trial. The following list of reported and/or potential AEs (Section 6.1) and the characteristics of an observed AE (Section 6.2) will determine whether the event requires expedited reporting **in addition** to routine reporting.

Adverse events will be monitored explicitly using a standardized adverse event form used in trials for psycho-active medications that will be reviewed by the study psychiatrists.

### **6.1** Expected Toxicities

Safety Profile

Gastrointestinal side effects of oral naltrexone (10-33%) include gastrointestinal symptoms such as nausea (>=10%), vomiting (>=3%), anorexia (<10%), constipation (<10%), and diarrhea (<10%). During controlled trials of oral naltrexone in alcohol dependence, approximately 5% of patients discontinued the drug because of nausea. CNS side effects of oral naltrexone include headache (>=7%), dizziness (4—9%), nervousness (>=4%), insomnia (>=3%), anxiety (>=2%), fatigue (>=4%), drowsiness (<=2%), increased energy (<10%), irritability (<10%), paranoia (<1%), restlessness (<1%), confusion (<1%), disorientation (<1%), hallucinations (<1%), nightmares (<1%), yawning (<1%), and hot flashes (<1%). Miscellaneous side effects include rash (<10%), increased thirst (<10%), and chills (<10%). Serious side effects of naltrexone (<1%) include hepatotoxicity (only reported at doses of 300mg/day or higher) and eosinophilic pneumonia (only reported with depot administration of naltrexone).

In controlled clinical trials of the extended-release injectable suspension of naltrexone, suicidal ideation, suicide attempts, or completed suicides occurred in 1% of patients and in no patients treated with placebo. In some cases, the suicidal thoughts or behavior occurred after study discontinuation but were in the context of an episode of depression that began while the patient was taking naltrexone. Although the incidence of adverse psychiatric events is expected to be considerably lower in the present study population as compared to populations of patients with alcohol and opioid dependence, depression and suicidal ideation will be systematically monitored during the present study using standardized self-report instruments.

Naltrexone blocks the effects of opioid analgesics and should not be used in patients who are currently on opioid analgesia, who have received opioids within the past 7 days (14 days for longer-acting opioids such as methadone), or who are expected to require opioid analgesia within the next 7 days. If opioids are required, the patient should stop naltrexone and wait 3 days before initiating opioids. If necessary, reversal of opioid blockade before the 3-day time period is possible to achieve, but should be done only under medical supervision, as higher doses may be required to achieve effective analgesia creating a risk of respiratory depression. Such supervision should occur in medical settings with the provision for respiratory support. This would include a hospital emergency department or intensive care unit.

Potential study participants will be strongly cautioned about unpleasant side effects of opioid withdrawal that may occur if they are on opioids at the time study drug is initiated. In addition, medication lists in LMR will be reviewed by study staff to verify the participant's self-report of opioid use.

Participants may use standard doses of acetaminophen, NSAIDs, or aspirin for analgesia during the study. Subjects on daily NSAIDs of >800mg ibuprofen daily (or the equivalent) will have LFTs one week after initiation of study drug. All participants will be instructed to report any symptoms of abdominal pain lasting more than a few days, white bowel movements, dark urine, or yellowing of their eyes. In the setting of these symptoms, liver function tests will be checked immediately.

Finally, if participants require opioid analgesia emergently during the course of the study, they will be taken off study. Study staff will notify the PI and QACT so that the treatment assignment (naltrexone or placebo) can be unblinded prior to initiating opioid analgesia. If the participant was assigned to naltrexone, the opioid analgesia will need to occur in a supervised medical setting, as above.

# 6.1.1 Adverse Events List(s) Adverse Event List(s) for naltrexone

| Common (10-33%) | Uncommon (1-10%) | Serious (<1%) |
|-----------------|------------------|-------------------------------|
| Nausea | Vomiting | Elevated liver function tests |
| | Anorexia | Suicidal ideation |
| | Diarrhea | |

| Constipation |
|------------------|
| Rash |
| Headache |
| Dizziness |
| Nervousness |
| Insomnia |
| Anxiety |
| Irritability |
| Increased thirst |

### **6.2** Adverse Event Characteristics

Reporting of adverse events:

All toxicities or adverse events occurring between the start of treatment and 30 days following the end of treatment will be recorded and graded as to severity and relationship to study drug. Any toxicity that is moderate or serious will be immediately reported by phone or email to the PI within 24 hours of discovery. All serious adverse reactions will be reported to the PI who will then notify the IRB.

A serious adverse reaction is defined as any of the following: life threatening; permanently disabling; requiring inpatient hospitalization or prolonging or hospitalization; death while on study treatment

A **moderate adverse reaction** is defined as the following: discomfort severe enough to cause interference with usual activities; persistent or requiring treatment

A **mild adverse reaction** is defined as the following: awareness of signs/symptoms, but easily tolerated; are of minor irritant type; causing no loss of time from normal activities; symptoms would not require medication or a medical evaluation; signs/symptoms are transient in nature

Preexisting medical conditions and symptoms related to known underlying diseases will not be recorded as adverse events unless they significantly worsen in severity during the course of the study.

Other than possible drug side effects, participants may also experience inconvenience and/or emotional distress, due to filling out instruments focusing on physical and emotional symptoms.

In case of subject distress, study psychiatrists can be contacted.

- CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP web site
  - $\underline{http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm}.$
- For expedited reporting purposes only:
  - AEs for the <u>agent(s)</u> that are listed above should be reported only if the adverse event

- varies in nature, intensity or frequency from the expected toxicity information which is provided.
- Other AEs for the <u>protocol</u> that do not require expedited reporting are outlined in the next section (Expedited Adverse Event Reporting) under the sub-heading of Protocol-Specific Expedited Adverse Event Reporting Exclusions.

### • **Attribution** of the AE:

- Definite The AE *is clearly related* to the study treatment.
- Probable The AE *is likely related* to the study treatment.
- Possible The AE *may be related* to the study treatment.
- Unlikely The AE *is doubtfully related* to the study treatment.
- Unrelated The AE *is clearly NOT related* to the study treatment.

## **6.3** Expedited Adverse Event Reporting

6.3.1 Investigators **must** report to the Overall PI any serious adverse event (SAE) that occurs after the initial dose of study treatment, during treatment, or within 30 days of the last dose of treatment on the local institutional SAE form.

### 6.3.2 <u>DF/HCC Expedited Reporting Guidelines</u>

Investigative sites within DF/HCC and DF/PCC will report SAEs directly to the DFCI Office for Human Research Studies (OHRS) per the DFCI IRB reporting policy.

### 6.3.3 Protocol-Specific Expedited Adverse Event Reporting Exclusions

N/A

# **6.4** Expedited Reporting to Hospital Risk Management

Participating investigators will report to their local Risk Management office any participant safety reports or sentinel events that require reporting according to institutional policy.

# **6.5** Routine Adverse Event Reporting

All Adverse Events must be reported in routine study data submissions to the Overall PI on the toxicity case report forms. AEs reported through expedited processes (e.g., reported to the IRB, FDA, etc.) must <u>also</u> be reported in routine study data submissions.

### 7. PHARMACEUTICAL INFORMATION

A list of the adverse events and potential risks associated with the investigational agent administered in this study can be found in Section 7.1.

### 7.1 Naltrexone

# 7.1.1 **Description**

Naltrexone (a pure opioid antagonist) is a cyclopropyl derivative of oxymorphone similar in structure to naloxone and nalorphine (a morphine derivative). The chemical name is N-Cyclopropylmethylnoroxymorphone and the formula is  $C_{20}H_{23}NO_4$ . The molecular weight is 341.40092. The NIM PubChem Compound ID is 5360515. Pharmacokinetic information follows below:

Duration: Oral: 25-50 mg: 24 hours

Absorption: Oral: Almost complete

Distribution: V<sub>d</sub>: ~1350 L; widely throughout the body but considerable interindividual

variation exists

Metabolism: Extensively metabolized via noncytochrome-mediated dehydrogenase conversion to 6-beta-naltrexol (primary metabolite) and related minor metabolites; glucuronide conjugates are also formed from naltrexone and its metabolites

Oral: Extensive first-pass effect

Protein binding: 21%

Bioavailability: Oral: Variable range (5% to 40%)

Half-life elimination: Oral: 4 hours; 6-beta-naltrexol: 13 hours; I.M.: naltrexone and 6-beta-

naltrexol: 5-10 days (dependent upon erosion of polymer)

Time to peak, serum: Oral: ~60 minutes; I.M.: Biphasic: ~2 hours (first peak), ~2-3 days

(second peak)

Excretion: Primarily urine (as metabolites and small amounts of unchanged drug)

Despite its hepatic metabolism, naltrexone does not interact with the cytochrome P450 enzyme system.

### 7.1.2 Form

Naltrexone is available generically from various manufacturers as a scored 50mg tablet (white or yellow in color).

### 7.1.3 Storage and Stability

Naltrexone hydrochloride tablets will be stored in well-closed containers at 15-30 degrees Celsius.

## 7.1.4 Compatibility

Not applicable for this study

# 7.1.5 Handling

No special considerations apply to handling for this study

### 7.1.6 Availability

The agent is commercially available from various manufacturers and will be purchased by the DFCI and MGH Research Pharmacies. Naltrexone will be purchased and billed to the study via established mechanisms at each site. It will be provided free of charge to participants.

# 7.1.7 Preparation

The DFCI and MGH Research Pharmacies will each purchase and over-encapsulate study medication and matching placebo per standard operating procedures of each site and provide the study drug supply for patients anticipated to go on the trial at the respective sites.

### 7.1.8 Administration

Orally dosed, once per day, in the morning with food.

### 7.1.9 **Ordering**

The agent will be obtained via commercial sources.

### 7.1.10 Accountability

As the responsible party designated by the investigator, the DFCI and MGH Research Pharmacies will maintain a careful record of the inventory and disposition of the agent using the NCI Drug Accountability Record Form (DARF) or another comparable drug accountability form. (See the NCI Investigator's Handbook for Procedures for Drug Accountability and Storage.)

### 7.1.11 Destruction and Return

At the end of the study, unused supplies of naltrexone will be destroyed according to institutional policies. Destruction will be documented according to the Drug Accountability Return Form.

### 8. BIOMARKER, CORRELATIVE, AND SPECIAL STUDIES

At the blood draw obtained for eligibility determination immediately prior to randomization, whole blood samples will be banked for analysis of OPRM1 (mu opioid receptor) genetic variants, specifically the Asn40Asp missense variant which has a frequency of 0.10-0.15 in Caucasians, 0.21 in Ashkenazi Jews, 0.25-0.45 in East Asians, and 0.14 in Hispanics.<sup>33</sup> The Asn40Asp variant has been shown to bind beta-endorphin approximately three times more tightly than the most common allelic form of the receptor,<sup>34</sup> and it has predicted good clinical response to naltrexone in alcohol and opioid dependence.<sup>33,35,36</sup>

Banked specimens will also be available for future exploratory examination of pro-inflammatory biomarkers such as expression-regulating polymorphisms in pro-inflammatory cytokine genes, which in recent studies have correlated with increased fatigue severity, depressive symptoms and memory complaints.<sup>37</sup>

Participants may opt out of specimen banking if they wish to do so.

# 9. STUDY CALENDARS

\*Note that study visits in both monitoring and intervention phase can be completed within 7 days of the scheduled date.

# Study measures, type of procedure, and study visit schedule **Monitoring Phase (6-week radiation therapy schedule)**

| Radiation TherapyBackground Information<br>Consent<br>Demographics/Patient<br>Characteristics Form<br>Clinical VariablesaXFatigue<br>FACIT-Fatigue Subscale<br>PGI-FSelf-report<br>Self-report<br>Self-reportXb<br>XbSleep<br>PSQI<br>ISI<br>ESS<br>Berlin QuestionnaireSelf-report<br>Self-report<br>Self-report<br>XbXb<br>XbOther Target Symptoms<br>GAD7<br>PHQ9Self-report<br>Self-report<br>Self-report<br>XbXc | |
|---|---|
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | |
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | |
| Characteristics Form<br>Clinical VariablesaTFatigue<br>FACIT-Fatigue Subscale<br>PGI-FSelf-report<br>Self-report $X^b$<br>Self-reportSleep<br>PSQI<br>ISI<br>ESS<br>Berlin QuestionnaireSelf-report<br>Self-report<br>Self-report<br>Self-report $X^b$<br>Self-report<br>$X^b$<br>Self-report<br>$X^b$ Other Target Symptoms<br>GAD7<br>PHQ9Self-report<br>Self-report<br>Self-report $X^b$<br>Self-report<br>$X^b$ | |
| Clinical Variablesa $X^a$ FatigueSelf-report $X^b$ FACIT-Fatigue SubscaleSelf-report $X^b$ PGI-FSelf-report $X^b$ SleepSelf-report $X^b$ PSQISelf-report $X^b$ ISISelf-report $X^b$ ESSSelf-report $X^b$ Berlin QuestionnaireSelf-report $X^b$ Other Target SymptomsSelf-report $X^b$ PHQ9Self-report $X^b$ | |
| FatigueSelf-report $X^b$ $X$ FACIT-Fatigue SubscaleSelf-report $X^b$ $X$ PGI-FSelf-report $X^b$ $X^b$ SleepSelf-report $X^b$ $X^b$ ISISelf-report $X^b$ $X^b$ ESSSelf-report $X^b$ $X^b$ Berlin QuestionnaireSelf-report $X^b$ $X^b$ Other Target SymptomsSelf-report $X^b$ $X^b$ PHQ9Self-report $X^b$ $X^c$ | |
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | |
| PGI-FSelf-report $X^b$ SleepSelf-report $X^b$ PSQISelf-report $X^b$ ISISelf-report $X^b$ ESSSelf-report $X^b$ Berlin QuestionnaireSelf-report $X^b$ Other Target Symptoms<br>GAD7Self-report $X^b$ PHQ9Self-report $X^b$ | |
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | X |
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | |
| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | |
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | |
| Berlin QuestionnaireSelf-report $X^b$ Other Target SymptomsSelf-report $X^b$ GAD7Self-report $X^b$ PHQ9Self-report $X^b$ $X^c$ | |
| GAD7 PHQ9 Self-report $X^b$ Self-report $X^c$ | |
| PHQ9 Self-report X <sup>b</sup> X <sup>c</sup> | |
| FACT-B/FACT-ES Self-report X <sup>b</sup> X <sup>c</sup> | |
| CPFQ Self-report X <sup>b</sup> | |
| PEG Self-report X <sup>b</sup> | |
| Safety monitoring | |
| Urine β-HCG | X |
| LFTs <sup>d</sup> | X |
| BUN/Creatinine d | X |
| Hematocrit <sup>d</sup> | X |
| TSH <sup>d</sup> | X |
| Subject Exit form (if | Xe |
| applicable) | |

a. Clinical Variables form completed once at end of radiation treatment for every patient in monitoring phase

b. baseline questionnaires to be completed within  $\leq$  21 days prior to, or within 3 days of starting radiation therapy, otherwise they need to be repeated.

c. During final week of RT, and 4 weeks after completion of RT

d. LFTs, BUN/Creatinine, Hematocrit will be accepted if drawn within 30 previous day; TSH within 6 months.

e. To be completed by study coordinator at time when patient is taken off-study for any reason. If patient continues on to Intervention Phase, this form will be completed when taken off intervention phase.

# Study measures, type of procedure, and study visit schedule **Monitoring Phase (Partial Breast Irradiation (PBI))**

| | Туре | Baseline Visit | Monitoring<br>Visits | Meets Fatigue<br>Eligibility<br>Threshold |
|---|---|---|---|---|
| <b>Background Information</b> | | | | |
| Consent | | X | | |
| Demographics/Patient | Self-report | X | | |
| Characteristics Form | | | | |
| Clinical Variables <sup>a</sup> | | | Xa | |
| Fatigue | | | | |
| FACIT-Fatigue Subscale | Self-report | $X^b$ | X <sup>c</sup> | X |
| PGI-F | Self-report | $X^b$ | | |
| Sleep | | | | |
| PSQI | Self-report | $X^b$ | | |
| ISI | Self-report | X <sup>b</sup> | | |
| ESS | Self-report | $X^b$ | | |
| Berlin Questionnaire | Self-report | $X^b$ | | |
| Other Target Symptoms | | | | |
| GAD7 | Self-report | $X^b$ | | |
| PHQ9 | Self-report | $X^b$ | $X^d$ | |
| FACT-B/FACT-ES | Self-report | $X^b$ | $X^d$ | |
| CPFQ | Self-report | $X^b$ | | |
| PEG | Self-report | X <sup>b</sup> | | |
| Safety monitoring | | | | |
| Urine $\beta$ -HCG | | | | X |
| LFTs <sup>e</sup> | | | | X |
| BUN/Creatinine <sup>e</sup> | | | | X |
| Hematocrit <sup>e</sup> | | | | X |
| TSH <sup>e</sup> | | | | X |
| Subject Exit form (if | | | | $X^{f}$ |
| applicable) | | | | |

a. Clinical Variables form completed once at end of radiation treatment for every patient in monitoring phase b. baseline questionnaires to be completed within  $\leq 21$  days prior to, or within 3 days of starting radiation therapy, otherwise they need to be repeated.

c. Complete once at baseline, once within one week after start of radiation, then once 4 weeks after completion of RT

d. Complete once at baseline, once within one week after start of radiation, then once while obtaining the final monitoring FACIT 4 weeks after end of RT

e. LFTs, BUN/Creatinine, Hematocrit will be accepted if drawn within 30 previous day; TSH within 6 months.

f. To be completed by study coordinator at time when patient is taken off-study for any reason. If patient continues on to Intervention Phase, this form will be completed when taken off intervention phase.

# Study measures, type of procedure, and study visit schedule **Monitoring Phase (Hypofractionation Radiation)**

| | Туре | Baseline Visit | Monitoring<br>Visits | Meets Fatigue<br>Eligibility<br>Threshold |
|---|---|---|---|---|
| <b>Background Information</b> | | | | |
| Consent | | X | | |
| Demographics/Patient | Self-report | X | | |
| Characteristics Form | | | | |
| Clinical Variables <sup>a</sup> | | | X <sup>a</sup> | |
| Fatigue | | | | |
| FACIT-Fatigue Subscale | Self-report | $X^b$ | X <sup>c</sup> | X |
| PGI-F | Self-report | $X^b$ | | |
| Sleep | | | | |
| PSQI | Self-report | $X^b$ | | |
| ISI | Self-report | $X^b$ | | |
| ESS | Self-report | $X^b$ | | |
| Berlin Questionnaire | Self-report | $X^b$ | | |
| Other Target Symptoms | | | | |
| GAD7 | Self-report | $X^b$ | | |
| PHQ9 | Self-report | $X^b$ | $X^d$ | |
| FACT-B/FACT-ES | Self-report | $X^b$ | $X^d$ | |
| CPFQ | Self-report | $X^b$ | | |
| PEG | Self-report | $X^b$ | | |
| Safety monitoring | | | | |
| Urine β-HCG | | | | X |
| LFTs <sup>e</sup> | | | | X |
| BUN/Creatinine <sup>e</sup> | | | | X |
| Hematocrit <sup>e</sup> | | | | X |
| TSH e | | | | X |
| Subject Exit form (if | | | | $X^{f}$ |
| applicable) | | | | |

a. Clinical Variables form completed once at end of radiation treatment for every patient in monitoring phase

b. baseline questionnaires to be completed within  $\leq$  21 days prior to, or within 3 days of starting radiation therapy, otherwise they need to be repeated.

c. Complete once at baseline, weekly during RT, then once 4 weeks after completion of RT

d. Complete once at baseline, once during the final week of RT, then once while obtaining the final monitoring FACIT 4 weeks after end of treatment

e. LFTs, BUN/Creatinine, Hematocrit will be accepted if drawn within 30 previous day; TSH within 6 months.

f. To be completed by study coordinator at time when patient is taken off-study for any reason. If patient continues on to Intervention Phase, this form will be completed when taken off intervention phase.

# Study measures, type of procedure, and study visit schedule Intervention Phase

| | Week 0<br>Randomi<br>zation<br>Visit | Week 1 Rx Visit (+/- 7 days) | Week 5 Rx<br>Visit (+/- 7<br>days) | Week 9 Follow-<br>up Visit (+/- 7<br>days) |
|---|---|---|---|---|
| <b>Background Information</b> | | | | |
| Consent | X | | | |
| Fatigue | | | | |
| FACIT-Fatigue Subscale | X | X | X | X |
| PGI-I | X | | X | |
| Sleep | | | | |
| PSQI | X | | X | |
| ISI | X | | X | |
| ESS | X | | X | |
| Berlin Questionnaire | | | X | |
| Other Target Symptoms | | | | |
| GAD7 | X | | X | |
| PHQ9 | X | | X | |
| FACT-B/FACT-ES | X | | X | |
| CPFQ | X | | X | |
| PEG | X | | X | |
| Safety monitoring | | | | |
| LFTs | | | X | |
| Concomitant medications | X | X | X | |
| Adverse Events assessment | | X | X | |
| Health status/life events review | | | | X |
| Dispense medication | X | X | | |
| Review medication diary | X | X | X | |
| Study Summary | | | | |
| Subject Exit form | | | | X <sup>a</sup> |
| Study Visit duration (min) | 40 | 15 | 40 | 15 |

a. To be completed by study coordinator at time when patient is taken off-study for any reason.

Effect measures listed in the Table of Procedures are described below. In addition to these effect measures, we will examine potential covariates that may play a role in the evolution of fatigue during breast radiotherapy. These include radiotherapy related characteristics such as breast volume; type of radiotherapy (e.g. fractionation schedule, number of fields, design of tangent fields [e.g. partial vs. full breast irradiation], boost dose [mini-tangents vs. electrons]. Exercise type/frequency and travel time to clinic will be assessed, as these parameters have correlated with radiotherapy-emergent fatigue in prior studies<sup>39</sup>. Finally, hematocrit will be measured at baseline.

The related symptom measure of obstructive sleep apnea will be evaluated via the Berlin Questionnaire and Epworth Sleepiness Scale:

Berlin Questionnaire (BQ): (Time: 2 minutes) The BQ will be done once at the beginning of the

study. It is an instrument used to identify patients at high risk for sleep apnea based on symptoms related to snoring and daytime sleepiness along with the presence of hypertension or obesity. It has been found to have high sensitivity and specificity in a primary care setting. <sup>40</sup>

<u>Epworth Sleepiness Scale (ESS):</u> (Time: 2 minutes) The ESS is a simple self-report scale of sleep propensity. The subject is asked to estimate the chances of dozing in each of 8 different situations on a scale of 0 to 3, with total scores ranging from 0 to 24. The ESS has been validated as a tool to differentiate normal subjects from those diagnosed with a sleep disorder. <sup>41</sup>

#### 10. MEASUREMENT OF EFFECT

The effect of naltrexone (and placebo in the control group) will be defined as a difference (in raw FACIT score) between the pre-randomization FACIT and the follow-up FACIT.

FACIT-fatigue subscale: This 13-item self-report scale measuring fatigue and functional impairment as a result of fatigue has been validated in cancer patients. It shows strong internal consistency (coefficient alpha range = 0.93-0.95) and test-retest reliability of  $0.82^{43}$ . The scale is reverse-scored and the range is 0 (maximum fatigue) - 52 (minimum fatigue). According to ICD-10 criteria, a score <= 34 indicates significant cancer related fatigue. A methodologically robust review of validated cancer-specific fatigue scales recommends the FACIT-fatigue subscale as the preferred outcome measure for research. 44

# 10.1 Other Response Parameters

Depression, anxiety, subjective cognitive function, sleep quality, insomnia, and quality of life outcome measures including pain will be assessed at study visits using the self-report measures listed below.

<u>GAD7</u>: (4 minutes) The Generalized Anxiety Disorder scale (GAD-7) is a 7-item self-report anxiety questionnaire which was initially validated in primary care populations; it has also been shown to be reliable and valid in the general population<sup>45</sup>. Of note, prior literature suggests that high baseline anxiety may be a risk factor for radiotherapy-emergent fatigue in breast cancer patients<sup>11</sup>

<u>Cognitive and Physical Functioning Scale</u> (CPFQ) (5 minutes): The CPFQ assesses both cognitive and physical functioning of individuals with mood and anxiety disorders. The CPFQ is a 7-item questionnaire that uses a 1-6 scale to measure impairment over the past month. The total score ranges from 6-42 points.

<u>Insomnia Severity Index (ISI)</u>: (4 minutes) The ISI is a subjective self-report assessment of sleep quality, restedness upon arising, daytime fatigue, attention/concentration and disturbances in relationships and mood. It is reliable and valid and has 7 items that use a 5-point Likert-style scale. Scores can range from 0 to 28. Of the 7 questionnaire items, 3 assess the severity of insomnia and 1 question each assesses satisfaction with current sleep pattern, sleep interference,

"noticeability" of sleeping problem to others, and concern about sleeping problems. 46

<u>Pittsburgh Sleep Quality Index (PSQI)</u>; (6 minutes) The PSQI is a widely used 19-item self-rated measure of sleep quality occurring during the one-month prior to assessment.<sup>47</sup> The PSQI has good test-retest reliability in healthy controls, depressed subjects, and sleep-disordered subjects.<sup>47</sup> The total PSQI score distinguishes healthy controls from individuals with depression and problems initiating and maintaining sleep.<sup>47</sup>

Functional Assessment of Cancer Therapy-Breast (FACT-B): (8 minutes) The FACT-B is a 37-item self-report questionnaire intended to assess quality of life in breast cancer patients. The measure is composed of 5 subscales: physical well being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and breast cancer related items (10 items). Subjects are asked to indicate how they have felt in the past 7 days on a 5-point Likert scale ranging from 0=Not at all to 4=Very much with higher scores indicating better quality of life. The FACT-B demonstrates good internal consistency (Cronbach's  $\alpha$ =0.88), good discriminative validity, and is sensitive to change.<sup>48</sup>

<u>Functional Assessment of Cancer Therapy-Endocrine Subscale (FACT-ES):</u> (4 minutes) Often used in combination with the FACT-B, the FACT-ES is intended to assess quality of life. Using the same 4 subscales of physical, social, emotional and functional well-being as the FACT-B, the FACT-ES contains an additional 19-item endocrine symptom subscale that assesses menopause symptoms. FACT-ES demonstrates good internal consistency, test-retest reliability, and sensitivity to change.<sup>49</sup>

<u>Patient Global Impression-Fatigue (PGI-Fatigue)</u>: (1 minute) This is a scale designed to assess global severity of fatigue and change in the patient's fatigue over time. This scale will be taken by the patient to assess severity of present fatigue and improvement relative to baseline state. It consists of 2 global subscales, severity of fatigue and global improvement. The clinician will determine the onset and duration for the symptoms as well as the impact of the symptoms on behavior and function in order to determine fatigue severity. The subscales are rated on 7-point scales with the range 0=not assessed to 7=Extremely ill. They have been found to be valid and reliable measures of fatigue and are validated with the CPFQ measure described above. <sup>50</sup>

<u>Patient Health Questionnaire (PHQ-9):</u> (3 minutes) The PHQ-9 is the self-administered form of the Primary Care Evaluation of Mental Disorders (PRIME-MD), a widely used instrument designed to screen for psychiatric illnesses in primary-care settings. The PHQ-9 is a 9-item self-report questionnaire that assesses mood, depressive symptoms, and suicidal ideation. It is used widely as a diagnostic screening tool for major depressive disorder, and has been found to be as good as longer clinician-rated interviews in a variety of settings. If any subject indicates suicidal ideation on the PHQ-9, she will be evaluated according to the suicide protocol described above in order to determine appropriate treatment and safety measures.<sup>51</sup>.

<u>PEG</u>: (1 minute). The PEG is an ultra-brief self-report scale measuring pain. It contains three items which assess average pain intensity (P), interference with enjoyable activities (E), and interference with general activity (G). It has been shown to have strong reliability, construct validity, and sensitivity to change in primary care and other ambulatory clinic patients.<sup>52</sup>

<u>Demographics/Patient Characteristics Form:</u> (3 minutes) This form will be completed by the patient to capture demographic, education, and prior health information.

<u>Clinical Variables</u>: Radiotherapy-related information to be completed by dosimetrist or physicist.

<u>Subject Exit Form</u>: This form will be completed by the study coordinator to capture summary of patient participation.

### 11. DATA REPORTING / REGULATORY REQUIREMENTS

Adverse event lists, guidelines, and instructions for AE reporting can be found in Section 7.0 (Adverse Events: List and Reporting Requirements).

# 11.1 Data Reporting

### 11.1.1 Method

Data is collected in an independent database created by the study team.

# 11.1.2 Responsibility for Data Submission

Investigative sites within DF/HCC or DF/PCC are responsible for collecting data variable within the study database.

# 11.2 Data Safety Monitoring

The DF/HCC Data and Safety Monitoring Board (DSMB) will review and monitor study progress, toxicity, safety and other data from this study. The board is chaired by a medical oncologist from outside of DF/HCC and has external and internal representation. Information that raises any questions about participant safety or protocol performance will be addressed by the Overall PI, statistician and study team. Should any major concerns arise, the DSMB will offer recommendations regarding whether or not to suspend the trial.

The DSMB will meet twice a year to review accrual, toxicity, response and reporting information. Information to be provided to the DSMB may include: participant accrual; treatment regimen information; adverse events and serious adverse events reported by category; summary of any deaths on study; audit results; and a summary provided by the study team. Other information (e.g. scans, laboratory values) will be provided upon request.

The study statistician, Andrzej Niemierko, will conduct the planned interim efficacy analysis. The PI will maintain oversight of administrative issues related to the analysis.

### 11.3 Multicenter Guidelines

N/A

### 11.4 Collaborative Agreements Language

N/A

### 12. STATISTICAL CONSIDERATIONS

Entry criteria of a drop of 10 points on FACIT-fatigue subscale was selected because a change of 10 points has been shown to constitute a clinically meaningful difference on this subscale<sup>53</sup>. The effect of naltrexone (and placebo in the control group) will be defined as a difference (in raw FACIT score) between the pre-randomization FACIT and the follow-up FACIT. FACIT-fatigue subscale scores are normally distributed in anemic and nonanemic cancer populations<sup>42</sup>, with a standard deviation of 10 points. Setting power as 0.8, and significance as 0.05, assuming a two-sided type I error, 122 patients per arm are required to detect a "difference of a difference" of at least 3.6 points on FACIT-fatigue. The 3.6 point difference was selected because it is the approximate mean of prior effect sizes utilizing FACIT-fatigue in clinical trials of erythropoeitin or darbopoeitin vs. placebo. Assuming a 20% drop-out rate, approximately 150 patients per arm will be randomized.

An interim analysis will be conducted on one occasion, after collecting data for the first 75 patients in each arm. This analysis will be conducted in light of several possibilities: 1) the observed benefit of naltrexone is so promising that it would be unethical not to use it for all eligible patients, 2) the observed rate of side effects/toxicity is too high, 3) futility –it appears to be unlikely that there is a clinically significant difference between the naltrexone and placebo arms. The Haybittle–Peto boundary rule (with 0.001 significance threshold) will be employed to determine whether the trial should be stopped early. The final analysis will still use the 0.05 threshold of significance.

Futility testing will also be performed on the primary outcome at a low level (one-sided alpha 0.0025) on one occasion (after the first 75 patients are enrolled).

# 12.1 Study Design/Endpoints

The study is a randomized placebo-controlled trial. The primary outcome measure will be change score on the FACIT-fatigue subscale from randomization to the end of the study. Exploratory endpoints include changes in sleep continuity (sleep efficiency, total sleep time, sleep latency), quality-of-life measures, depression, anxiety, and subjective cognitive function.

Analysis of both the primary and exploratory endpoints will be by modified intention to treat. The mITT analysis (for both primary and exploratory endpoints) will be a per-protocol analysis; only patients who complete the entire trial according to the protocol will be counted towards the final results.

# 12.2 Sample Size/Accrual Rate

Sample size for the intervention phase of the study is 150 patients per arm randomized to treatment. Assuming a 4 year study duration, and 2 study sites, we will randomize 1-2
participants per study site every 2 weeks (~75 randomized participants / year). The sample size for the monitoring phase of the study is not fixed, but using a conservative estimate of 30% for radiation treatment-emergent fatigue, we will need to screen 3-6 participants per study site per 2 weeks (~225 screened participants / year).

### 12.3 Stratification Factors

Patients will be stratified according to whether or not they received chemotherapy.

### 12.4 Analysis of Secondary Endpoints

Secondary (exploratory) endpoints (changes in sleep continuity (sleep efficiency, total sleep time, sleep latency), quality-of-life measures, depression, anxiety, and subjective cognitive function) will be analyzed by modified intention to treat. Since no pre-existing data describes the magnitude of associations of our exploratory outcomes with naltrexone use in this population, we are unable to speculate on the statistical power required to detect an effect. Any relevant associations and their statistical significances will be calculated using descriptive statistics. In addition, radiation therapy status (currently receiving RT vs. recently completed RT) will be included as a covariate in the multivariate analysis.

### 12.5 Reporting and Exclusions

### 12.5.1 Evaluation of Toxicity

All participants will be evaluable for toxicity from the time of their first treatment. Some patients may tolerate the 25mg dose but develop toxicity after the dose is increased to 50mg. Hence, drug dose can be decreased from 50mg to 25mg in the setting of moderate to severe adverse events by CTCAE judged to be definitely or probably related to study drug.

Study drug (either at the 25mg or 50mg dose) can also be held for up to three days and then restarted in setting of moderate or severe adverse events by CTCAE if these events are judged to be possible, unlikely or unrelated to study drug. If the drug must be held for more than three days, the participant will need to come off the study.

### 12.5.2 Evaluation of Response

All of the participants who meet the eligibility criteria, consent to randomization, and complete the entire treatment protocol will be included in the main analysis of effect.

For all dropouts, we will use an off-study form in order to obtain information about the reasons for not completing the study. We will use this information for post-hoc analyses to lessen the chance of bias due to missing data.

### 13. PUBLICATION PLAN

The results will be made public within 24 months of the end of data collection. A report is planned to be published in a peer-reviewed journal and that initial release may be an abstract that meets the requirements of the International Committee of Medical Journal Editors. A full report of the outcomes will be made public no later than three years after the end of data collection.

### APPENDIX A INFORMATION ON POSSIBLE DRUG INTERACTIONS

### Information on Possible Interactions with Other Agents for Patients and Their Caregivers and Non-Study Healthcare Team

| The participant | is enrolled on a clinical trial using the |
|---|---|
| experimental agent [naltrexone]. This clinical tria | l is sponsored by the National Cancer |
| Institute. This form is addressed to the participant, | but includes important information for |
| others who care for this participant. | |

Naltrexone blocks the effects of opioid containing medications, including pain medications such as Percocet, Vicodin, Oxycodone, Oxycontin, Dilaudid, Fentanyl, and Methadone; as well as Codeine and Loperamide. Because of this, it is very important to tell your study doctors about all of your medicine before you start this study. It is also very important to tell them if you stop taking any regular medicine, or if you start taking a new medicine while you take part in this study. When you talk about your medicine with your study doctor, include medicine you buy without a prescription at the drug store (over-the-counter remedy), or herbal supplements such as St. John's wort.

Many health care prescribers can write prescriptions. You must also tell your other prescribers (doctors, physicians' assistants or nurse practitioners) that you are taking part in a clinical trial. **Bring this paper with you and keep the attached information card in your wallet**. These are the things that you and they need to know:

You will be asked to avoid taking any opioid containing medication which will not work because naltrexone blocks the effects of opioids, including pain relief. Furthermore, the use of narcotics will require that you drop out of the study. Naltrexone does not interfere with the effectiveness of non-narcotic pain relievers (e.g., acetaminophen [Tylenol], ibuprofen, and local or general anesthesia). If you need an opioid medication for a medical procedure (e.g., surgery) that can be scheduled in advance, your medication can be discontinued prior to your surgery. If you are scheduled for a surgical procedure, you must inform us so that we can let your treating physician, dentist, and/or anesthesiologist know that you may be taking naltrexone, an opiate blocker.

You will be asked to carry a medication card which will, in case of emergency, alert the medical personnel treating you that you may be taking naltrexone, an opioid blocker. This card, which should be kept on you at all times, will include appropriate drug information and precautions. A second card will be provided which must be given to a family member to keep at home for reference purposes.

| INFORMATION | ON ON POSSIBLE DRUG INTERACTIONS |
|---|---|
| You are enrolled on | a clinical trial using the agent |
| · | This clinical trial is sponsored by the NCI. |
| 442770 | blocks the effects of opioid containing |
| medications. Becau | se of this, it is very important to: |
| ➤ Tell your doctors | if you stop taking regular medicine or if you start |
| taking a new medici | ine. 3 ANCER |
| > Tell all of your pr | escribers (doctor, physicians' assistant, nurse |
| practitioner, and ph | armacist) that you are taking part in a clinical |
| trial. | |
| Check with your | doctor or pharmacist whenever you need to us $ angle 2$ |
| an over-the-counter | r medicine or herbal supplement. |

| > You must notify your doctors that you are on naltrexone if you |
|------------------------------------------------------------------|
| require surgery, or if you develop pain requiring management |
| with opioid containing medications |
| > Your study doctor's name is |
| and can be contacted at |

### References

- 1. Zucca AC, Boyes AW, Linden W, Girgis A. All's well that ends well? Quality of life and physical symptom clusters in long-term cancer survivors across cancer types. Journal of pain and symptom management 2012;43:720-31.
- 2. Goldstein D, Bennett B, Friedlander M, Davenport T, Hickie I, Lloyd A. Fatigue states after cancer treatment occur both in association with, and independent of, mood disorder: a longitudinal study. BMC cancer 2006;6:240.
- 3. Alvarez J, Meyer FL, Granoff DL, Lundy A. The Effect of EEG Biofeedback on Reducing Postcancer Cognitive Impairment. Integrative cancer therapies 2013.
- 4. Sanford SD, Beaumont JL, Butt Z, Sweet JJ, Cella D, Wagner LI. Prospective Longitudinal Evaluation of a Symptom Cluster in Breast Cancer. Journal of pain and symptom management 2013.
- 5. Kangas M, Bovbjerg DH, Montgomery GH. Cancer-related fatigue: a systematic and meta-analytic review of non-pharmacological therapies for cancer patients. Psychological bulletin 2008;134:700-41.
- 6. Minton O, Richardson A, Sharpe M, Hotopf M, Stone P. A systematic review and meta-analysis of the pharmacological treatment of cancer-related fatigue. Journal of the National Cancer Institute 2008;100:1155-66.
- 7. Jean-Pierre P, Morrow GR, Roscoe JA, et al. A phase 3 randomized, placebo-controlled, double-blind, clinical trial of the effect of modafinil on cancer-related fatigue among 631 patients receiving chemotherapy: a University of Rochester Cancer Center Community Clinical Oncology Program Research base study. Cancer 2010;116:3513-20.
- 8. Monk JP, Phillips G, Waite R, et al. Assessment of tumor necrosis factor alpha blockade as an intervention to improve tolerability of dose-intensive chemotherapy in cancer patients. Journal of clinical oncology: official journal of the American Society of Clinical Oncology 2006;24:1852-9.
- 9. Bower JE, Ganz PA, Aziz N. Altered cortisol response to psychologic stress in breast cancer survivors with persistent fatigue. Psychosomatic medicine 2005;67:277-80.
- 10. Spiegel D, Giese-Davis J, Taylor CB, Kraemer H. Stress sensitivity in metastatic breast cancer: analysis of hypothalamic-pituitary-adrenal axis function. Psychoneuroendocrinology 2006;31:1231-44.
- 11. Courtier N, Gambling T, Enright S, Barrett-Lee P, Abraham J, Mason MD. A prognostic tool to predict fatigue in women with early-stage breast cancer undergoing radiotherapy. Breast 2013;22:504-9.
- 12. Manir KS, Bhadra K, Kumar G, Manna A, Patra NB, Sarkar SK. Fatigue in breast cancer patients on adjuvant treatment: course and prevalence. Indian journal of palliative care 2012;18:109-16.
- 13. Geinitz H, Zimmermann FB, Stoll P, et al. Fatigue, serum cytokine levels, and blood cell counts during radiotherapy of patients with breast cancer. International journal of radiation oncology, biology, physics 2001;51:691-8.
- 14. Greenberg DB, Sawicka J, Eisenthal S, Ross D. Fatigue syndrome due to localized radiation. Journal of pain and symptom management 1992;7:38-45.
- 15. Irvine DM, Vincent L, Graydon JE, Bubela N. Fatigue in women with breast cancer receiving radiation therapy. Cancer nursing 1998;21:127-35.
- 16. Donovan KA, Jacobsen PB, Andrykowski MA, et al. Course of fatigue in women

- receiving chemotherapy and/or radiotherapy for early stage breast cancer. Journal of pain and symptom management 2004;28:373-80.
- 17. Taunk NK, Haffty BG, Chen S, et al. Comparison of radiation-induced fatigue across 3 different radiotherapeutic methods for early stage breast cancer. Cancer 2011;117:4116-24.
- 18. Reidunsdatter RJ, Albrektsen G, Hjermstad MJ, Rannestad T, Oldervoll LM, Lundgren S. One-year course of fatigue after post-operative radiotherapy in Norwegian breast cancer patients--comparison to general population. Acta Oncol 2013;52:239-48.
- 19. Huang YP, Lin MT, Chen JS, Wu PY. Naltrexone protects against hypotension, hyperthermia, and beta-endorphin overproduction during heatstroke in the rat. Journal of pharmacological sciences 2005;97:519-24.
- 20. Strassman RJ, Appenzeller O, Lewy AJ, Qualls CR, Peake GT. Increase in plasma melatonin, beta-endorphin, and cortisol after a 28.5-mile mountain race: relationship to performance and lack of effect of naltrexone. The Journal of clinical endocrinology and metabolism 1989;69:540-5.
- 21. Cazzullo AG, Musetti MC, Musetti L, Bajo S, Sacerdote P, Panerai A. Beta-endorphin levels in peripheral blood mononuclear cells and long-term naltrexone treatment in autistic children. European neuropsychopharmacology: the journal of the European College of Neuropsychopharmacology 1999;9:361-6.
- 22. Krupitsky E, Nunes EV, Ling W, Illeperuma A, Gastfriend DR, Silverman BL. Injectable extended-release naltrexone for opioid dependence: a double-blind, placebo-controlled, multicentre randomised trial. Lancet 2011;377:1506-13.
- 23. Anton RF, O'Malley SS, Ciraulo DA, et al. Combined pharmacotherapies and behavioral interventions for alcohol dependence: the COMBINE study: a randomized controlled trial. JAMA: the journal of the American Medical Association 2006;295:2003-17.
- 24. Greenway FL, Fujioka K, Plodkowski RA, et al. Effect of naltrexone plus bupropion on weight loss in overweight and obese adults (COR-I): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet 2010;376:595-605.
- 25. Epperson CN, Toll B, Wu R, et al. Exploring the impact of gender and reproductive status on outcomes in a randomized clinical trial of naltrexone augmentation of nicotine patch. Drug and alcohol dependence 2010;112:1-8.
- 26. Anton RF. Naltrexone for the management of alcohol dependence. The New England journal of medicine 2008;359:715-21.
- 27. Ciraulo DA, Dong Q, Silverman BL, Gastfriend DR, Pettinati HM. Early treatment response in alcohol dependence with extended-release naltrexone. The Journal of clinical psychiatry 2008;69:190-5.
- 28. Hofman M, Ryan JL, Figueroa-Moseley CD, Jean-Pierre P, Morrow GR. Cancer-related fatigue: the scale of the problem. The oncologist 2007;12 Suppl 1:4-10.
- 29. Schwartz AL, Nail LM, Chen S, et al. Fatigue patterns observed in patients receiving chemotherapy and radiotherapy. Cancer investigation 2000;18:11-9.
- 30. Cui R, Widlund HR, Feige E, et al. Central role of p53 in the suntan response and pathologic hyperpigmentation. Cell 2007;128:853-64.
- 31. Mickley GA, Stevens KE, Burrows JM, White GA, Gibbs GL. Morphine tolerance offers protection from radiogenic performance deficits. Radiation research 1983;93:381-7.
- 32. Lowe SW, Bodis S, McClatchey A, et al. p53 status and the efficacy of cancer therapy in vivo. Science 1994;266:807-10.
- 33. Oroszi G, Anton RF, O'Malley S, et al. OPRM1 Asn40Asp predicts response to

- naltrexone treatment: a haplotype-based approach. Alcoholism, clinical and experimental research 2009;33:383-93.
- 34. Bond C, LaForge KS, Tian M, et al. Single-nucleotide polymorphism in the human mu opioid receptor gene alters beta-endorphin binding and activity: possible implications for opiate addiction. Proceedings of the National Academy of Sciences of the United States of America 1998;95:9608-13.
- 35. Anton RF, Oroszi G, O'Malley S, et al. An evaluation of mu-opioid receptor (OPRM1) as a predictor of naltrexone response in the treatment of alcohol dependence: results from the Combined Pharmacotherapies and Behavioral Interventions for Alcohol Dependence (COMBINE) study. Archives of general psychiatry 2008;65:135-44.
- 36. Chamorro AJ, Marcos M, Miron-Canelo JA, Pastor I, Gonzalez-Sarmiento R, Laso FJ. Association of micro-opioid receptor (OPRM1) gene polymorphism with response to naltrexone in alcohol dependence: a systematic review and meta-analysis. Addiction biology 2012;17:505-12.
- 37. Bower JE, Ganz PA, Irwin MR, Castellon S, Arevalo J, Cole SW. Cytokine genetic variations and fatigue among patients with breast cancer. Journal of clinical oncology: official journal of the American Society of Clinical Oncology 2013;31:1656-61.
- 38. Kim SW, Grant JE, Adson DE, Remmel RP. A preliminary report on possible naltrexone and nonsteroidal analgesic interactions. Journal of clinical psychopharmacology 2001;21:632-4.
- 39. Purcell A, Fleming J, Bennett S, McGuane K, Burmeister B, Haines T. A multidimensional examination of correlates of fatigue during radiotherapy. Cancer 2010;116:529-37.
- 40. Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Annals of internal medicine 1999;131:485-91.
- 41. Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep 1991;14:540-5.
- 42. Cella D, Lai JS, Chang CH, Peterman A, Slavin M. Fatigue in cancer patients compared with fatigue in the general United States population. Cancer 2002;94:528-38.
- 43. Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. Journal of pain and symptom management 1997;13:63-74.
- 44. Minton O, Stone P. A systematic review of the scales used for the measurement of cancer-related fatigue (CRF). Annals of oncology: official journal of the European Society for Medical Oncology / ESMO 2009;20:17-25.
- 45. Lowe B, Decker O, Muller S, et al. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Medical care 2008;46:266-74.
- 46. Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Medicine 2001;2:297-307.
- 47. Buysse DJ, Reynolds CFd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res 1989;28:193-213.
- 48. Brady MJ, Cella DF, Mo F, et al. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. Journal of clinical oncology: official journal of the American Society of Clinical Oncology 1997;15:974-86.

- 49. Fallowfield LJ, Leaity SK, Howell A, Benson S, Cella D. Assessment of quality of life in women undergoing hormonal therapy for breast cancer: validation of an endocrine symptom subscale for the FACT-B. Breast cancer research and treatment 1999;55:189-99.
- 50. Targum SD, Hassman H, Pinho M, Fava M. Development of a clinical global impression scale for fatigue. Journal of psychiatric research 2012;46:370-4.
- 51. Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med 2007;22:1596-602.
- 52. Krebs EE, Lorenz KA, Bair MJ, et al. Development and initial validation of the PEG, a three-item scale assessing pain intensity and interference. Journal of general internal medicine 2009;24:733-8.
- 53. Reddy S, Bruera E, Pace E, Zhang K, Reyes-Gibby CC. Clinically important improvement in the intensity of fatigue in patients with advanced cancer. Journal of palliative medicine 2007;10:1068-75.

### **OTHER MEDICATIONS TAKEN**

If you take a daily medication (prescribed or otherwise), please use one line per drug and indicate the start and stop dates under the "Date(s) Taken" section (i.e., 6/2/09 - 6/5/09).

### Study Participant Self-Administration Study Drug Diary

Dana-Farber/Harvard Cancer Center

| Participant Identifier: | Protocol #: 14-056 | Your MD Phone | Your RN Phone | STUDY DRUG INSTRUCTIONS: | Study Drug: Naltrexone/Placebo | How Much: Your dose is | <b>How Often:</b> You will take each dose once a day | When: You should take your dose in the morning with food | SPECIAL INSTRUCTIONS: | If you miss or vomit a dose, you may retake the drug within 8 hours of missing or vomiting that dose. | ) | Capsules must be swallowed whole | As a reminder, please bring any unused study drug, all empty | containers, and this drug diary to your next clinic visit. | | | | SYMPTOMS/SIDE EFFECTS | Please record any side effects experienced during this cycle. | Include the date the particular symptom started and when it |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Reason Taken | | | | | | | | | | | | | | | returned: | | | | | |
| Dates Taken | | | | | | | | | | Date | | USE ONLY | | Date Returned: | # pills/caps/tabs returned: | 1,000 | Ken: | | | |
| Dose | | | | | | | | | | | | FOR STUDY TEAM USE ONLY | | | | the second creek | nave been ta | | | |
| Drug Name | | | | | | | | | | Study Participant Initials | | FOR STUI | Staff Initials: | Date Dispensed: | # pills/caps/tabs dispensed: | 4 11:042 404 2404/2000/211:04 H | # pilis/caps/tabs tnat snouid nave been taken: | Discrepancy Notes: | | |

ended. Please evaluate the severity of the symptom according to

the following scale:

### DOSING TOG

Naltrexone RCT for Treatment-Emergent Fatigue in Patients Receiving Radiation

Therapy for Breast Cancer

Cycle: \_\_\_\_ For each AM dose take:

Please indicate the date, time, amount taken and any comments.

Mild: Awareness of sign or symptom; easily tolerated and did not affect ability to perform normal daily activities. Symptom did not require medication or therapeutic intervention.

**Moderate:** Significant discomfort which interfered with ability to perform normal daily activities. Symptom was easily resolved with at home medication or simple therapeutic intervention.

Please Note: The severity should reflect the most severe level Start Date End Date | Severity normal daily activities. Symptom required new medication Severe: Marked discomfort with an inability to carry out and/or therapeutic intervention in order to resolve. experienced during the time period. Symptom vomited pill Comments Time and Amount Taken For each AM dose take: Naltrexone/Placebo 8 am - 1 6/1/2009 Date Cycle: \_ Day 3 Day 5 Day 6 Day 7 Day 4 Day 2 Day 1 Ex:

Please indicate the date, time, amount taken and any comments.

vomited pill Comments Time and Amount Taken 8 am -6/1/2009 Date Day 10 Day 12 Day 13 Day 14 Day 17 Day 15 Day 11 Day 16 Day 8 Day 9 Ex:

| Day 18 | Day 19 | Day 20 | Day 21 | Day 22 | Day 23 | Day 24 | Day 25 | Day 26 | Day 27 | Day 28 | Day 29 | Day 30 | Day 31 | Day 32 | Day 33 | Day 34 | Day 35 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

| Patient ID: | Date: |
|-------------|-------|
| Visit: | |

### The PEG

| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
|---|---|---|---|---|---|---|---|---|---|---|
| Noţ | oain | | | | | | | | | Pain as bad as<br>you can imagin |
| | | | est des<br>ent of l | | s how, | during | g the p | ast we | ek, pa | in has interfered |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | s not | | | | | | | | | Completely<br>interferes |
| inter | rrere | | | | | | | | | |
| Wh<br>ith y | at nun | eneral | activit | у? | - | • | | | | in has interfered |
| ith y | at nun | eneral | activit | у? | s how, | • | | | ek, pa | in has interfered |

| Patient signature/initials: |
|-----------------------------|
| Date: |

### SAFTEE (1)

Below is a list of complaints people sometimes have. Please read each and circle the number corresponding to how much you have been bothered by that problem in the past week:

| 1 = not at all | 2 = a little bit | 3 = moderately | 4 = quite a bit | 5 = extremely |
|---|---|---|---|---|
| i iiotataii | _ ~ | o illoadlately | i quito a sit | o oxeronion |

| Head: | | | | | |
|---------------------------------------|----------|--------|---------|---|----|
| 1. headaches | 1 | 2 | 3 | 4 | 5 |
| 2. dizziness or faintness | 1 | 2 | 3 | 4 | 5 |
| 3. loss of consciousness | 1 | 2 | 3 | 4 | 5 |
| 4. seizures | 1 | 2 | 3 | 4 | 5 |
| Any other problems with your head | l (pleas | se spe | ecify): | | |
| 5. | 1 | 2 | 3 | 4 | 5 |
| 6. | 1 | 2 | 3 | 4 | 5 |
| Eyes: | | | | | |
| 7. eye irritation | 1 | 2 | 3 | 4 | 5 |
| 8. swelling | 1 | 2 | 3 | 4 | 5 |
| 9. blurred vision | 1 | 2 | 3 | 4 | 5 |
| 10. double vision | 1 | 2 | 3 | 4 | 5 |
| 11. poor vision | 1 | 2 | 3 | 4 | 5 |
| 12. light bothering your eyes | 1 | 2 | 3 | 4 | 5 |
| Any other problems with your eyes | (pleas | se spe | cify): | | |
| 13. | 1 | 2 | 3 | 4 | 5 |
| 14. | 1 | 2 | 3 | 4 | 5 |
| Ears: | | | | | |
| 15. earache | 1 | 2 | 3 | 4 | 5 |
| 16. discharge | 1 | 2 | 3 | 4 | 5 |
| 17. trouble hearing | 1 | 2 | 3 | 4 | 5 |
| 18. ringing or whistling or other noi | se in e | ars | | | |
| 1 2 3 4 5 | | | | | |
| Any other problems with your ears | | | | | |
| <u>19.</u> | 1 | 2 | 3 | 4 | 5 |
| 20. | 1 | 2 | 3 | 4 | 5- |
| Mouth and Teeth: | | | | | |
| 21. sores in your mouth | 1 | 2 | 3 | 4 | 5 |
| 22. dry mouth | 1 | 2 | 3 | 4 | 5 |
| 23. too much saliva | 1 | 2 | 3 | 4 | 5 |
| 24. swollen or sore tongue | 1 | 2 | 3 | 4 | 5 |
| 25. bleeding gums | 1 | 2 | 3 | 4 | 5 |
| 26. dental problems | 1 | 2 | 3 | 4 | 5 |

| Any other problems with your mouth | or to | oth (r | معدما | enac | if <sub>V</sub> )· |
|---|---|---|---|---|---|
| 27. | 1 | 2 | 3 | 4 | 5 |
| 28. | 1 | 2 | 3 | 4 | 5 |
| Nose and Throat: | | | | | |
| 29. nasal congestion | 1 | 2 | 3 | 4 | 5 |
| 30. nose bleeds | 1 | 2 | 3 | 4 | 5 |
| 31. sore throat | 1 | 2 | 3 | 4 | 5 |
| 32. laryngitis | 1 | 2 | 3 | 4 | 5 |
| 33. difficulty swallowing | 1 | 2 | 3 | 4 | 5 |
| Any other problems with your nose of | r thr | oat (pi | ease | specii | fy): |
| 34. | 1 | 2 | 3 | 4 | 5 |
| 35. | 1 | 2 | 3 | 4 | 5 |
| Chest: | | | | | |
| 36. chest pain | 1 | 2 | 3 | 4 | 5 |
| 37. shortness of breath | 1 | 2 | 3 | 4 | 5 |
| 38. wheezing | 1 | 2 | 3 | 4 | 5 |
| 39. coughing | 1 | 2 | 3 | 4 | 5 |
| 40. breast or nipple pain or discharge | e 1 | 2 | 3 | 4 | 5 |
| 41. breast tenderness | 1 | 2 | 3 | 4 | 5 |
| Any other trouble with your chest (ple | ease | speci | fy): | | |
| 42. | 1 | 2 | 3 | 4 | 5 |
| 43. | 1 | 2 | 3 | 4 | 5 |
| Heart: | | | | | |
| 44. rapid heart rate | 1 | 2 | 3 | 4 | 5 |
| 45. irregular heart beat | 1 | 2 | 3 | 4 | 5 |
| Any other trouble with your heart (ple | ease | speci | fy): | | |
| 46. | 1 | 2 | 3 | 4 | 5 |
| 47. | 1 | 2 | 3 | 4 | 5 |
| Stomach and Abdomen: | | | | | |
| 48. stomach / abdominal discomfort | 1 | 2 | 3 | 4 | 5 |
| 49. nausea | 1 | 2 | 3 | 4 | 5 |
| 50. vomiting | 1 | 2 | 3 | 4 | 5 |
| 51. heartburn | 1 | 2 | 3 | 4 | 5 |

### SAFTEE (2)

Below is a list of complaints people sometimes have. Please read each and circle the number corresponding to how much you have been bothered by that problem in the past week:

| 1 = not at all | 2 = a little bit | 3 = moderately | 4 = quite a bit | 5 = extremely |
|---|---|---|---|---|

| Any other trouble with stomach or all | bdom | en (pl | ease | specii | fy): |
|---|---|---|---|---|---|
| 52. | 1 | 2 | 3 | 4 | 5 |
| 53. | 1 | 2 | 3 | 4 | 5 |
| Bowel: | | | | | |
| 54. diarrhea | 1 | 2 | 3 | 4 | 5 |
| 55. constipation | 1 | 2 | 3 | 4 | 5 |
| 56. gas | 1 | 2 | 3 | 4 | 5 |
| 57. change in color of stools | 1 | 2 | 3 | 4 | 5 |
| 58. hemorrhoids | 1 | 2 | 3 | 4 | 5 |
| 59. painful bowel movements | 1 | 2 | 3 | 4 | 5 |
| Any other changes in your bowel mo | ovem | ents ( <sub>l</sub> | please | spec | cify): |
| 60. | 1 | 2 | 3 | 4 | 5 |
| 61. | 1 | 2 | 3 | 4 | 5 |
| Appetite: | | | | | |
| 62. appetite increase | 1 | 2 | 3 | 4 | 5 |
| 63. appetite decrease | 1 | 2 | 3 | 4 | 5 |
| 64. weight gain | 1 | 2 | 3 | 4 | 5 |
| 65. weight loss | 1 | 2 | 3 | 4 | 5 |
| 66. bad taste or change in taste | 1 | 2 | 3 | 4 | 5 |
| 67. increased thirst | 1 | 2 | 3 | 4 | 5 |
| Any other change in appetite (please | e spe | cify): | | | |
| 68. | 1 | 2 | 3 | 4 | 5 |
| 69. | 1 | 2 | 3 | 4 | 5 |
| Urination: | | | | | |
| 70. painful urination | 1 | 2 | 3 | 4 | 5 |
| 71. burning sensation with urination | 1 | 2 | 3 | 4 | 5 |
| 72. difficulty in starting to urinate | 1 | 2 | 3 | 4 | 5 |
| 73. decrease in force of urinary stream | am | | | | |
| 1 2 3 4 5 | | | | | |
| 74. more frequent urination | 1 | 2 | 3 | 4 | 5 |
| 75. change in color of urine 1 2 3 4 | | | 5 | | |
| Any other problems with urination (p | lease | spec | ify): | | |
| 76. | 1 | 2 | 3 | 4 | 5 |
| 77. | 1 | 2 | 3 | 4 | 5 |

| ely 4 = quite a bit 5 = extreme | ely | | | | |
|---|---|---|---|---|---|
| FEMALES: | | | | | |
| 78. menstrual irregularity | 1 | 2 | 3 | 4 | 5 |
| 79. cramps | 1 | 2 | 3 | 4 | 5 |
| 80. heavy bleeding | 1 | 2 | 3 | 4 | 5 |
| 81. spotting | 1 | 2 | 3 | 4 | 5 |
| 82. tension | 1 | 2 | 3 | 4 | 5 |
| 83. hot flashes | 1 | 2 | 3 | 4 | 5 |
| 84. lengthening of menstrual period | | | | | |
| | 1 | 2 | 3 | 4 | 5 |
| 85. shortening of menstrual period | | | | | |
| | 1 | 2 | 3 | 4 | 5 |
| Any other problems with menstrual | period | l (plea | se sp | ecify). | |
| 86. | 1 | 2 | 3 | 4 | 5 |
| 87. | 1 | 2 | 3 | 4 | 5 |
| Genital and Sexual Functioning: | | | | | |
| 88. discomfort in genitals | 1 | 2 | 3 | 4 | 5 |
| 89. swelling of or discharge from ge | nitals | | | | |
| | 1 | 2 | 3 | 4 | 5 |
| 90. decrease in interest in sex | 1 | 2 | 3 | 4 | 5 |
| 91. increase in interest in sex | 1 | 2 | 3 | 4 | 5 |
| 92. delayed orgasm or inability to re | ach o | rgasm | ) | | |
| | 1 | 2 | 3 | 4 | 5 |
| 93. MALES: difficulty achieving or r | nainta | ining a | an ere | ection | |
| | 1 | 2 | 3 | 4 | 5 |
| Any other problems with genitals or | sexua | al func | tionin | g (ple | ase |
| specify): | | | | | |
| 94. | 1 | 2 | 3 | 4 | 5 |
| 95. | 1 | 2 | 3 | 4 | 5 |

### SAFTEE (3)

Below is a list of complaints people sometimes have. Please read each and circle the number corresponding to how much you have been bothered by that problem in the past week:

1 = not at all 2 = a little bit 3 = moderately 4 = quite a bit 5 = extremely

| Muscles, Bones and Joints: | | | | | |
|---|---|---|---|---|---|
| 96. aches, pains in muscles, bones | or joi | nts | | | |
| | 1 | 2 | 3 | 4 | 5 |
| 97. swelling in legs or arms | 1 | 2 | 3 | 4 | 5 |
| 98. tingling or numbness in hands o | r feet | | | | |
| | 1 | 2 | 3 | 4 | 5 |
| Any other trouble with your muscles | , bon | es, or | joints | (plea | se |
| specify): | | | | | |
| 99. | 1 | 2 | 3 | 4 | 5 |
| 100. | 1 | 2 | 3 | 4 | 5 |
| Walking and Moving: | | | | | _ |
| 101. feeling unsteady on your feet | 1 | 2 | 3 | 4 | 5 |
| 102. trouble with starting to move | 1 | 2 | 3 | 4 | 5 |
| 103. controlling unwanted bodily mo | veme | ents | | | |
| | 1 | 2 | 3 | 4 | 5 |
| 104. feeling restless or like you can | not st | ay stil | Ì | | _ |
| | 1 | 2 | 3 | 4 | 5 |
| 105. shaking | 1 | 2 | 3 | 4 | 5 |
| 106. feeling still or rigid | 1 | 2 | 3 | 4 | 5 |
| Any other difficulty with walking or n | novin | g (plea | ase sp | pecify) | ): |
| 107. | 1 | 2 | 3 | 4 | 5 |
| 108. | 1 | 2 | 3 | 4 | 5 |
| Scalp and Skin: | | | | | |
| 109. rashes, itching, or irritation | 1 | 2 | 3 | 4 | 5 |
| 110. bruising | 1 | 2 | 3 | 4 | 5 |
| 111. increased irritation in sunlight | 1 | 2 | 3 | 4 | 5 |
| 112. sweating a lot | 1 | 2 | 3 | 4 | 5 |
| Any other trouble with your scalp or | skin | (pleas | e spe | cify): | |
| 113. | 1 | 2 | 3 | 4 | 5 |
| 114. | 1 | 2 | 3 | 4 | 5 |

| Other Areas: | | | | | |
|---|---|---|---|---|---|
| 115. fever or chills | 1 | 2 | 3 | 4 | 5 |
| 116. feeling tired or fatigued | 1 | 2 | 3 | 4 | 5 |
| 117. too much energy | 1 | 2 | 3 | 4 | 5 |
| 118. jumpiness or feeling jittery | 1 | 2 | 3 | 4 | 5 |
| 119. feeling excited, overactive, or e | elated | j | | | |
| | 1 | 2 | 3 | 4 | 5 |
| 120. problems falling asleep | 1 | 2 | 3 | 4 | 5 |
| 121. problems staying asleep | 1 | 2 | 3 | 4 | 5 |
| 122. waking up too early | 1 | 2 | 3 | 4 | 5 |
| 123. sleeping too much | 1 | 2 | 3 | 4 | 5 |
| 124. feeling drowsy during the day | 1 | 2 | 3 | 4 | 5 |
| 125. trouble thinking, concentrating | , or re | ememl | bering | | |
| | 1 | 2 | 3 | 4 | 5 |
| 126. feeling down, depressed or blu | ıe1 | 2 | 3 | 4 | 5 |
| 127. feeling anxious | 1 | 2 | 3 | 4 | 5 |
| 128. irritability | 1 | 2 | 3 | 4 | 5 |
| Any other problems with your thinking | ng, m | ood, e | energy | , or o | ther |
| aspects of your health (please spec | ify): | | | | |
| 129. | 1 | 2 | 3 | 4 | 5 |
| 130. | 1 | 2 | 3 | 4 | 5 |
| 131. | 1 | 2 | 3 | 4 | 5 |
| 132. | 1 | 2 | 3 | 4 | 5 |

Protocol: 2009-P-001557 Impact of HF on Sleep and Mood

PI: Hadine Joffe, MD

| Subject ID: | | | | _ |
|-------------|-------|----|---|---|
| Visit #: | Date: | /_ | / | |

### PITTSBURG SLEEP QUALITY INDEX

| | - | | | <del></del> |
|---|---|---|---|---|
| Th | | | | ng the past month <u>only</u> . |
| | Your answers should indicate the most accurate replay for the <u>majority</u> of days and nights in the past month. Please answer all questions. | | | |
| 1. | During the past | month, what time hav | e you usually gone to | bed at night? |
| | | BED T | TME | |
| 2. | During the past month, how long (in minutes) has it usually taken you to fall asleep each night? | | | |
| | | NUMBER OF | MINUTES | |
| 3. | During the past | month, what time hav | e you usually gotten | up in the morning? |
| | | GETTING | UP TIME | |
| 4. | | month, how many hou<br>that the number of ho | | I you get at night? (This<br>.) |
| | | HOURS OF SLEE | P PER NIGHT | <u></u> |
| | r each of the ren<br>questions. | naining questions, c | heck the one best r | esponse. Please answer |
| 5. | During the past | month, how often hav | e you had trouble sle | eping because you |
| a) | Cannot get to | o sleep within 30 min | utes | |
| | t during<br>st month | Less than once a week | Once or twice a week | Three or more times a week |
| b) | | he middle of the night | | times a week |
| , | · | _ | , | |
| | | Less than once a week | | Three or more times a week |
| c) | Have to get | up to use the bathroo | m | |
| | t during<br>st month | Less than once a week | Once or twice a week | Three or more times a week |

Protocol: 2009-P-001557 Impact of HF on Sleep and Mood PI: Hadine Joffe, MD

| ubject ID: | | | |
|------------|-------|---|---|
| /isit#: | Date: | / | / |

| d) Cannot breatl | ne comfortably | | |
|---|---|---|---|
| Not during past month | Less than once a week | Once or twice a week | Three or more times a week |
| e) Cough or sno | re loudly | | |
| | Less than once a week | | Three or more times a week |
| f) Feel too cold | | | |
| Not during past month | Less than once a week | Once or twice a week | Three or more times a week |
| g) Feel too hot | | | |
| • | Less than once a week | | Three or more times a week |
| h) Had bad drea | ims | | |
| | Less than once a week | Once or twice a week | Three or more times a week |
| i) Have pain | | | |
| • | Less than once a week | | Three or more times a week |
| j) Other reason | (s), please describe | | |
| Not during past month | Less than once a week | Once or twice a week | Three or more times a week |
| 6. During the past n | nonth, how would you r | rate your sleep quality | overall? |
| | Very good | | |
| | Fairly good | | |
| | Fairly bad | | |
| | Very bad | | |

Reprinted by permission of the author, Daniel J. Buysse, M.D.

| Protocol: 2009-P-Impact of HF on SPI: Hadine Joffe, I | Sleep and | l Mood | | S | ubject ID 'isit #: | :<br>Date: | / | _/ |
|---|---|---|---|---|---|---|---|---|
| 7. During the prescribed or ' | | onth, how often have<br>ne counter")? | you taken medi | cine to I | nelp you | ı sleep | | |
| Not during past month | | Less than once a week | Once or twice a week | | Three c | | | |
| | | onth, how often have<br>ging in social activity′ | | staying | ı awake | while dri | ving, | |
| | | Less than once a week | | | Three c | | | |
| | | onth, how much of a post things done? | problem has it b | een for | you to k | eep up | | |
| | No pro | blem at all | | | | | | |
| | Only a | very slight problem | | | | | | |
| | Somew | hat of a problem | | | | | | |
| , | Very ba | ad | | | | | | |
| Patient Initia | ıls/Sigi | nature: | | | | | | |
| Date | | | | | | | | |

| Patient ID: |
|-------------|
| Date: |
| Visit#: |

### PHQ-9 — Nine Symptom Checklist

| 1. | Over the last 2 weeks, how often have you been bothered by any of the following problems? Read each item carefully, and circle your response. | | | |
|---|---|---|---|---|
| | a. Little interest or<br>Not at all | r pleasure in doing thin<br>Several days | ngs<br>More than half the days | Nearly every day |
| | b. Feeling down, o | lepressed, or hopeless<br>Several days | More than half the days | Nearly every day |
| | c. Trouble falling Not at all | asleep, staying asleep,<br>Several days | or sleeping too much More than half the days | Nearly every day |
| | d. Feeling tired or<br>Not at all | having little energy<br>Several days | More than half the days | Nearly every day |
| | e. Poor appetite or<br>Not at all | overeating<br>Several days | More than half the days | Nearly every day |
| | f. Feeling bad abo<br>yourself or your fa<br>Not at all | • | nt you are a failure, or feeling t More than half the days | hat you have let Nearly every day |
| | g. Trouble concen | trating on things such Several days | as reading the newspaper or w More than half the days | ratching television Nearly every day |
| | | | ner people could have noticed.<br>nd a lot more than usual<br>More than half the days | Or being so fidgety or<br>Nearly every day |
| | i. Thinking that yo | ou would be better off of Several days | dead or that you want to hurt y More than half the days | ourself in some way<br>Nearly every day |
| 2. | • | • • | questionnaire so far, how diffic<br>rk, take care of things at home | |
| | Not Difficult at | all Somewhat Diffi | icult Very Difficult | Extremely Difficult |
| | | ure: | | |
| Da | te: | | | |

| Patient | : ID: |
|----------|-------|
| Date: | |
| Visit #: | |

### PATIENT GLOBAL IMPRESSIONS: SEVERITY OF FATIGUE

Targum and Fava © Massachusetts General Hospital

Symptoms of fatigue may include effects on:

### Your physical wellbeing:

Low or decreased energy, tiredness, decreased physical endurance or ability to sustain physical activity, general weakness, heaviness in the arms or legs, general heaviness, slowness or sluggishness, sleepiness, increased effort with physical tasks.

### Your mood state:

Decreased motivation or interest, decreased effort or initiative.

### Your cognitive abilities:

Decreased concentration, decreased attention, slowed thinking, reduced mental sharpness.

Within the past week, how troublesome (disturbing or distressing) have the identified symptoms of fatigue been for you?

### CIRCLE THE NUMBER CORRESPONDING TO YOUR RATING

| 1 | Normal, no symptoms of | No symptoms of fatigue have been present in the |
|---|---|---|
| | fatigue | past seven days |
| 2 | Borderline symptoms | There may have been subtle symptoms of fatigue |
| | | but there was no meaningful impact on your |
| | | behavior or function |
| 3 | Mild fatigue | There have been some clear symptoms of fatigue |
| | | but they may have cause minimal, if any, |
| | | emotional distress or difficulty for you in social |
| | | or occupational situations |
| 4 | Moderate fatigue | There have been overt (definite) symptoms of |
| | | fatigue causing noticeable, but modest, functional |
| | | difficulties (impairment) or distress for you; |
| | | These symptoms are interfering with (but not |

| | | stopping) social, educational, or occupational |
|---|---|---|
| | | function |
| 5 | Marked fatigue | There have been intrusive symptoms of fatigue |
| | | that distinctly impair social or occupational |
| | | activities or function and/or cause high levels of |
| | | distress; The functional interference due to these |
| | | symptoms is obvious to others |
| 6 | Severe fatigue | The symptoms of fatigue are very distressing to |
| | | you and are disrupting behavior or function in |
| | | multiple domains of function (social, occupation, |
| | | school) |
| 7 | Extreme fatigue | Symptoms of fatigue are drastically interfering |
| | | in many life functions; You may be unable to |
| | | work or attend school |

| Patient Initials/Signature: | <br> |
|-----------------------------|------|
| Date: | |

| Patient | i ID: |
|----------|-------|
| Date: | |
| Visit #: | |

### PATIENT GLOBAL IMPRESSIONS-IMPROVEMENT

Targum and Fava © Massachusetts General Hospital

Rate total improvement of fatigue within the past week whether or not it is due entirely to drug treatment

Compared to how you felt previously, how much have you changed over the past week?

### CIRCLE THE NUMBER CORRESPONDING TO YOUR RATING

| 1 | Very much improved | Nearly all better; good level of functioning; |
|---|---|---|
| | | Minimal symptoms of fatigue if any at all; |
| | | This level represents a very substantial change |
| | | from the baseline assessment |
| 2 | Much improved | Notably better with significant reduction of symptoms; |
| | | Increase in the level of functioning but some symptoms |
| | | of fatigue may remain |
| 3 | Minimally improved | Slightly better; There may be only a modest change in |
| | | symptoms of fatigue or functional capacity |
| 4 | No change | Symptoms of fatigue remain essentially unchanged |
| 5 | Minimally worse | Slightly worse but may not be clinically meaningful; |
| | | There may be only a modest worsening of symptoms or |
| | | functioning |
| 6 | Much worse | Notably worse with significant increase of symptoms of |
| | | fatigue; Associated decrease in the level of functioning |
| 7 | Very much worse | Severe exacerbation of symptoms and profound impact |
| | | on behavior and/or functioning |

| Patient Initials/Signature: | |
|-----------------------------|---|
| Date: | _ |

| Patient ID: _ | <br> |
|---------------|------|
| Date: | <br> |
| Visit #: | |

Table 1. Massachusetts General Hospital CPFQ

| 1 | 2 | st/enthusiasm been over | 4 | 5 | 6 |
|---|---|---|---|---|---|
| greater | normal | minimally | moderately | markedly | totally |
| than normal | 1102111111 | diminished | diminished | diminished | absent |
| (b) How has you | r wakefulness/alert | ness been over the past 1 | nonth? | | - |
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater | normal | minimally | moderately | markedly | totally |
| than normal | | diminished | diminished | diminished | absent |
| (c) How has your | energy been over t | he past month? | | | |
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater | normal | minimally | moderately | markedly | totally |
| than normal | | diminished | diminished | diminished | absent |
| (d) How has you | r ability to focus/su | stain attention been ove | er the past month? | | ======================================= |
| 1 | 2 | 3 | 4Visit: | Dat <b>§:</b> / / | 6 |
| greater | normal | minimally | moderately | markedly | totally |
| than normal | | diminished | diminished | diminished | absent |
| (e) How has your | ability to rememb | er/recall information be | en over the past mon | th? | |
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater | normal | minimally | moderately | markedly | totally |
| than normal | | diminished | diminished | diminished | absent |
| (f) How has your | ability to find wor | ds been over the past me | onth? | | |
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater | normal | minimally | moderately | markedly | totally |
| than normal | | diminished | diminished | diminished | absent |
| | sharpness/mental | acuity been over the pa | st month? | | |
| (g) How has your | | | 4 | 5 | 6 |
| (g) How has you<br>1 | 2 | 3 | 4 | 5 | 0 |
| (g) How has your<br>1<br>greater | 2<br>normal | 3<br>minimally | moderately | markedly | totally |

Please answer all questions by *circling* the *correct answer* or the answer which seems the most *appropriate* to you (consider 'normal' the time in your life prior to the past month when you were most satisfied with your cognitive and physical functioning). Copyright: Massachusetts General Hospital.

| Patient Initials/Signature: |
|-----------------------------|
| Date: |

| Patient I | D: |
|-----------|----|
| Date: | |
| Visit#: | |

### **Insomnia Severity Index**

For each question, please CIRCLE the number that best describes your answer.

Please rate the CURRENT (i.e. LAST 2 WEEKS) SEVERITY of your insomnia problem(s).

| Insomnia Problem | None | Mild | Moderate | Severe | Very Severe |
|---|---|---|---|---|---|
| 1. Difficulty falling asleep | 0 | 1 | 2 | 3 | 4 |
| 2. Difficulty staying asleep | 0 | 1 | 2 | 3 | 4 |
| 3. Problems waking up too early | 0 | 1 | 2 | 3 | 4 |

| 3. Problems waking up too early | | | 0 | 1 | 2 | 3 | |
|---|---|---|---|---|---|---|---|
| 4. How SATISFIED/DI | SSATISFIEI | o are you wi | th your CUR | RENT sleep | pattern? | | |
| Very Satisfied | Satisfied | | ely Satisfied | | • | Dissatisfied | |
| 0 | 1 | | 2 | 3 | • | 4 | |
| 5. How NOTICEABLE your life? Not at all | to others do | you think yo | our sleep pro | blem is in ter | ms of impairi | ing the quality | y of |
| Noticeable | A Little | Somewh | at Muc | eh Verv | Much Notic | eable | |
| 0 | 1 | 2 | 3 | - | 4 | cuote | |
| 6. How WORRIED/DIS<br>Not at all<br>Worried<br>0 | STRESSED a A Little 1 | re you abou<br>Somewh | • | | em? Much Worr 4 | ied | |
| 7. To what extent do yo daytime fatigue, mood, CURRENTLY? Not at all Interfering 0 | | | k/daily chore | es, concentrat | | , mood, etc.) | e.g. |
| v | | 2 | | | · | | |

| Patient Initials/Signature: _ |
|-------------------------------|
| Date: |

| Subject ID: | | | |
|-------------|-------|---|-------|
| Visit #: | Date: | / | <br>/ |

### **Generalized Anxiety Disorder – 7 questions**

Instructions: for each question below, please circle the number of the statement that best matches how you feel

How often during the past 2 weeks have you felt bothered by:

- 1. Feeling nervous, anxious, or on edge?
  - 0 = not at all
  - 1 = several days
  - 2 = more than half the days
  - 3 = nearly everyday
- 2. Not being able to stop or control worrying?
  - 0 = not at all
  - 1 = several days
  - 2 = more than half the days
  - 3 = nearly everyday
- 3. Worrying too much about different things?
  - 0 = not at all
  - 1 = several days
  - 2 = more than half the days
  - 3 = nearly everyday
- 4. Trouble relaxing?
  - 0 = not at all
  - 1 = several days
  - 2 = more than half the days
  - 3 = nearly everyday

- 5. Being so restless that it is hard to sit still?
  - 0 = not at all
  - 1 =several days
  - 2 = more than half the days
  - 3 = nearly everyday
- 6. Becoming easily annoyed or irritable?
  - 0 = not at all
  - 1 = several days
  - 2 = more than half the days
  - 3 = nearly everyday
- 7. Feeling afraid as if something awful might happen?
  - 0 = not at all
  - 1 =several days
  - 2 = more than half the days
  - 3 = nearly everyday

If you checked off any problems, how difficult have these problems made it for you to do your work, take care of things at home, or get along with other people?

### (Please circle one option below)

- Not difficult at all
- Somewhat difficult
- Very difficult
- Extremely difficult

| Patient Initials/Signature: |
|-----------------------------|
| Date: |

### Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (Version 4)

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the past 7 days.

| | | Not At All | A Little Bit | Somewhat | Quite a Bit | Very Much |
|---|---|---|---|---|---|---|
| 1 | I feel fatigued | 0 | 1 | 2 | 3 | 4 |
| 2 | I feel weak all over | 0 | 1 | 2 | 3 | 4 |
| 3 | I feel listless ("washed out") | 0 | 1 | 2 | 3 | 4 |
| 4 | I feel tired | 0 | 1 | 2 | 3 | 4 |
| 5 | I have trouble <u>starting</u> things<br>because I am tired | 0 | 1 | 2 | 3 | 4 |
| 6 | I have trouble <u>finishing</u> things<br>because I am tired | 0 | 1 | 2 | 3 | 4 |
| 7 | I have energy | 0 | 1 | 2 | 3 | 4 |
| 8 | I am able to do my usual activities | 0 | 1 | 2 | 3 | 4 |
| 9 | I need to sleep during the day | 0 | 1 | 2 | 3 | 4 |
| 10 | I am too tired to eat | 0 | 1 | 2 | 3 | 4 |
| 11 | I need help doing my usual activities | 0 | 1 | 2 | 3 | 4 |
| 12 | I am frustrated by being too tired<br>to do the things I want to do | 0 | 1 | 2 | 3 | 4 |
| 13 | I have to limit my social activity<br>because I am tired | 0 | 1 | 2 | 3 | 4 |

Scoring: Items are scored as follows: 4=Not At All; 3=A Little Bit; 2=Somewhat; 1=Quite A Bit; 0=Very Much, EXCEPT items #7 and #8 which are reversed scored. Score range 0-52. A score of less than 30 indicates severe fatigue. The higher the score, the better the quality of life.

| Item Number | Reverse Item? | | Item Response | Item Score |
|-------------|---------------|----|---------------|------------|
| 1 | 4 | - | * | = |
| 2 | 4 | - | | = |
| 3 | 4 | - | | = |
| 4 | 4 | - | | = |
| 5 | 4 | 92 | | = |
| 6 | 4 | - | | = |
| 7 | 0 | + | | = |
| 8 | 0 | + | | = |
| 9 | 4 | - | | |
| 10 | 4 | - | | = |
| 11 | 4 | - | | = |
| 12 | 4 | 2 | | = |
| 13 | 4 | | | # |

| Sum individual it | em scores: | | | |
|---|---|---|---|---|
| Multiply by 13: | | | | |
| Divide by number | r of items answered: | === | | |
| contribite on the time booker | | | <br> | . 0 . 1 1. |

For guidelines on handling missing data and scoring options, please refer to the Administration and Scoring Guidelines on-line at www.facit.org.

Source: Webster, K., Cella, D., & Yost, K. (2003). The functional assessment of chronic illness therapy (FACIT) measurement system: properties, applications and interpretation. *Health and Quality of Life Outcomes*, 1(79), 1-7.

Reprinted with permission from: http://www.facit.org/FACITOrg/Questionnaires



A series provided by The Hartford Institute for Genatric Nursing, New York University, College of Nursing

| Patient I | D: |
|-----------|----|
| Date: | |
| Visit#: | |

### **FACT-B (Version 4)**

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the past 7 days.

| | | PHYSICAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|---|
| | GP1 | I have a lack of energy | 0 | 1 | 2 | 3 | 4 |
| | GP2 | I have nausea | 0 | 1 | 2 | 3 | 4 |
| | GP3 | Because of my physical condition, I have trouble meeting the needs of my family | 0 | 1 | 2 | 3 | 4 |
| | GP4 | I have pain | 0 | 1 | 2 | 3 | 4 |
| | GP5 | I am bothered by side effects of treatment | 0 | 1 | 2 | 3 | 4 |
| | GP6 | I feel ill | 0 | 1 | 2 | 3 | 4 |
| | GP7 | I am forced to spend time in bed | 0 | 1 | 2 | 3 | 4 |
| ĺ | | SOCIAL/FAMILY WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
| | GS1 | I feel close to my friends | 0 | 1 | 2 | 3 | 4 |
| | GS2 | I get emotional support from my family | 0 | 1 | 2 | 3 | 4 |
| | GS3 | I get support from my friends | 0 | 1 | 2 | 3 | 4 |
| | GS4 | My family has accepted my illness | 0 | 1 | 2 | 3 | 4 |
| | GS5 | I am satisfied with family communication about my illness | 0 | 1 | 2 | 3 | 4 |
| | GS6 | I feel close to my partner (or the person who is my main support) | 0 | 1 | 2 | 3 | 4 |
| | Q1 | Regardless of your current level of sexual activity, please answer the following question. If you prefer not to answer it, please mark this box and go to the next section. | | | | | |
| | GS7 | I am satisfied with my sex life | 0 | 1 | 2 | 3 | 4 |

| Patient I | D: |
|-----------|----|
| Date: | |
| Visit#: | |

### FACT-B (Version 4)

Please circle or mark one number per line to indicate your response as it applies to the past 7 days.

| | EMOTIONAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| GE1 | I feel sad | 0 | 1 | 2 | 3 | 4 |
| GE2 | I am satisfied with how I am coping with my illness | 0 | 1 | 2 | 3 | 4 |
| GE3 | I am losing hope in the fight against my illness | 0 | 1 | 2 | 3 | 4 |
| GE4 | I feel nervous | 0 | 1 | 2 | 3 | 4 |
| GE5 | I worry about dying | 0 | 1 | 2 | 3 | 4 |
| GE6 | I worry that my condition will get worse | 0 | 1 | 2 | 3 | 4 |
| | FUNCTIONAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
| GF1 | FUNCTIONAL WELL-BEING I am able to work (include work at home) | | | | - | • |
| GF1 | | at all | bit | what | a bit | much |
| | I am able to work (include work at home) | at all | <b>bit</b> | what | a bit | much 4 |
| GF2 | I am able to work (include work at home) | 0<br>0<br>0 | <b>bit</b> 1 1 | <b>what</b> 2 2 | 3 3 3 | <b>4</b> 4 |
| GF2<br>GF3 | I am able to work (include work at home) | 0<br>0<br>0<br>0 | bit 1 1 1 | 2<br>2<br>2 | 3 3 3 | 4<br>4<br>4 |
| GF2<br>GF3<br>GF4 | I am able to work (include work at home) | 0<br>0<br>0<br>0 | bit 1 1 1 1 | 2<br>2<br>2<br>2 | 3 3 3 3 3 | 4<br>4<br>4<br>4 |

| Patient I | D: |
|-----------|----|
| Date: | |
| Visit#: | |

### FACT-B (Version 4)

Please circle or mark one number per line to indicate your response as it applies to the past 7 days.

| | ADDITIONAL CONCERNS | Not at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| В1 | I have been short of breath | 0 | 1 | 2 | 3 | 4 |
| B2 | I am self-conscious about the way I dress | 0 | 1 | 2 | 3 | 4 |
| В3 | One or both of my arms are swollen or tender | 0 | 1 | 2 | 3 | 4 |
| B4 | I feel sexually attractive | 0 | 1 | 2 | 3 | 4 |
| В5 | I am bothered by hair loss | 0 | 1 | 2 | 3 | 4 |
| В6 | I worry that other members of my family might | | | | | |
| | someday get the same illness I have | 0 | 1 | 2 | 3 | 4 |
| В7 | I worry about the effect of stress on my illness | 0 | 1 | 2 | 3 | 4 |
| В8 | I am bothered by a change in weight | 0 | 1 | 2 | 3 | 4 |
| В9 | I am able to feel like a woman | 0 | 1 | 2 | 3 | 4 |
| P2 | I have certain parts of my body where I experience pain | 0 | 1 | 2 | 3 | 4 |

| Patient Initials/Signature: | |
|-----------------------------|---|
| Date: | _ |

| Patient ID: _ | |
|---------------|----------|
| Date: | |
| /isit#: | <u> </u> |

### **FACT-ES** (Version 4)

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the past 7 days.

| ĺ | | PHYSICAL WELL-BEING | Not<br>at all | A little<br>bit | Some<br>-what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|---|
| | GP1 | I have a lack of energy | 0 | 1 | 2 | 3 | 4 |
| | GP2 | I have nausea | 0 | 1 | 2 | 3 | 4 |
| | GP3 | Because of my physical condition, I have trouble meeting the needs of my family | 0 | 1 | 2 | 3 | 4 |
| | GP4 | I have pain | 0 | 1 | 2 | 3 | 4 |
| | GP5 | I am bothered by side effects of treatment | 0 | 1 | 2 | 3 | 4 |
| | GP6 | I feel ill | 0 | 1 | 2 | 3 | 4 |
| | GP7 | I am forced to spend time in bed | 0 | 1 | 2 | 3 | 4 |
| | | SOCIAL/FAMILY WELL-BEING | Not<br>at all | A little<br>bit | Some<br>-what | Quite<br>a bit | Very<br>much |
| | GS1 | I feel close to my friends | 0 | 1 | 2 | 3 | 4 |
| | GS2 | I get emotional support from my family | 0 | 1 | 2 | 3 | 4 |
| | GS3 | I get support from my friends | 0 | 1 | 2 | 3 | 4 |
| | GS4 | My family has accepted my illness | 0 | 1 | 2 | 3 | 4 |
| | GS5 | I am satisfied with family communication about my illness | 0 | 1 | 2 | 3 | 4 |
| | GS6 | I feel close to my partner (or the person who is my main support) | 0 | 1 | 2 | 3 | 4 |
| | Q1 | Regardless of your current level of sexual activity, please answer the following question. If you prefer not to answer it, please mark this box and go to the next section. | | | | | |
| | GS7 | I am satisfied with my sex life | 0 | 1 | 2 | 3 | 4 |

| Patient ID: |
|-------------|
| Date: |
| Visit#: |

### **FACT-ES** (Version 4)

Please circle or mark one number per line to indicate your response as it applies to the past 7 days.

| | EMOTIONAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| GE1 | I feel sad | 0 | 1 | 2 | 3 | 4 |
| GE2 | I am satisfied with how I am coping with my illness | 0 | 1 | 2 | 3 | 4 |
| GE3 | I am losing hope in the fight against my illness | 0 | 1 | 2 | 3 | 4 |
| GE4 | I feel nervous | 0 | 1 | 2 | 3 | 4 |
| GE5 | I worry about dying | 0 | 1 | 2 | 3 | 4 |
| GE6 | I worry that my condition will get worse | 0 | 1 | 2 | 3 | 4 |
| | FUNCTIONAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
| GF1 | FUNCTIONAL WELL-BEING I am able to work (include work at home) | | | | - | • |
| GF1 | | at all | bit | what | a bit | much |
| | I am able to work (include work at home) | o<br>0 | <b>bit</b><br>1 | what | a bit | much 4 |
| GF2 | I am able to work (include work at home) | 0<br>0<br>0 | <b>bit</b> 1 1 | <b>what</b> 2 2 | 3 3 | <b>4</b> 4 |
| GF2<br>GF3 | I am able to work (include work at home) | 0<br>0<br>0<br>0 | bit 1 1 1 | 2<br>2<br>2 | 3 3 3 | 4<br>4<br>4 |
| GF2<br>GF3<br>GF4 | I am able to work (include work at home) | 0<br>0<br>0<br>0 | bit 1 1 1 1 | 2<br>2<br>2<br>2 | 3 3 3 3 3 | 4<br>4<br>4<br>4 |

| Patient | ID: |
|---------|-----|
| Date: | |
| Visit#: | |

### FACT-ES (Version 4)

Please circle or mark one number per line to indicate your response as it applies to the past 7 days.

| Ī | | ADDITIONAL CONCERNS | Not<br>at all | A<br>little | Some<br>-what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|---|
| | ES1 | I have hot flashes | 0 | 1 | 2 | 3 | 4 |
| | ES2 | I have cold sweats | 0 | 1 | 2 | 3 | 4 |
| | ES3 | I have night sweats | 0 | 1 | 2 | 3 | 4 |
| | ES4 | I have vaginal discharge | 0 | 1 | 2 | 3 | 4 |
| | ES5 | I have vaginal itching/irritation | 0 | 1 | 2 | 3 | 4 |
| | ES6 | I have vaginal bleeding or spotting | 0 | 1 | 2 | 3 | 4 |
| | ES7 | I have vaginal dryness | 0 | 1 | 2 | 3 | 4 |
| | ES8 | I have pain or discomfort with intercourse | 0 | 1 | 2 | 3 | 4 |
| | ES9 | I have lost interest in sex | 0 | 1 | 2 | 3 | 4 |
| | ES10 | I have gained weight | 0 | 1 | 2 | 3 | 4 |
| | An9 | I feel lightheaded (dizzy) | 0 | 1 | 2 | 3 | 4 |
| | O2 | I have been vomiting | 0 | 1 | 2 | 3 | 4 |
| | C5 | I have diarrhea (diarrhoea) | 0 | 1 | 2 | 3 | 4 |
| | An10 | I get headaches | 0 | 1 | 2 | 3 | 4 |
| | Tax1 | I feel bloated | 0 | 1 | 2 | 3 | 4 |
| | ES11 | I have breast sensitivity/tenderness | 0 | 1 | 2 | 3 | 4 |
| | ES12 | I have mood swings | 0 | 1 | 2 | 3 | 4 |
| | ES13 | I am irritable | 0 | 1 | 2 | 3 | 4 |
| | BRM<br>1 | I have pain in my joints | 0 | 1 | 2 | 3 | 4 |

| Patient Initials/Signature: |
|-----------------------------|

Date:

| Patient ID | <b>:</b> |
|------------|----------|
| Date: | |
| Visit#: | |

### **Epworth Sleepiness Scale**

How likely are you to doze off or fall asleep in the situations described below, in contrast to feeling just tired?

This refers to your usual way of life in recent times.

Even if you haven't done some of these things recently try to work out how they would have affected you.

Use the following scale to choose the most appropriate number for each situation:-

- 0 =Would never doze
- 1 = Slight chance of dozing
- $2 = \underline{\text{Moderate}}$  chance of dozing
- $3 = \underline{\text{High}}$  chance of dozing

| Sitting and reading |
|-------------------------------------------------------------------|
| Watahing TV |
| Watching TV |
| Sitting, inactive in a public place (e.g. a theatre or a meeting) |
| As a passenger in a car for an hour without a break |
| Lying down to rest in the afternoon when circumstances permit |
| Sitting and talking to someone |
| Sitting quietly after a lunch without alcohol |
| In a car, while stopped for a few minutes in the traffic |

Patient Initials/Signature:

Date: \_\_\_\_\_

| Patient ID:<br>Date: | |
|---|---|
| Visit#: | |
| BERLIN QUESTIONNAIRE | |
| Height (m) Weight (kg) Age | Male / Female |
| Please choose the correct response to each question. | |
| CATEGORY 1 | CATEGORY 2 |
| 1. Do you snore? | 6. How often do you feel tired or fatigued after |
| ☐ a. Yes | your sleep? |
| □ b. No | a. Nearly every day |
| ☐ c. Don't know | b. 3-4 times a week |
| If you snore: | c. 1-2 times a week |
| y you shore. | d. 1-2 times a month |
| 2. Your snoring is: | e. Never or nearly never |
| <ul><li>a. Slightly louder than breathing</li><li>b. As loud as talking</li></ul> | 7. During your waking time, do you feel tired, fatigued or not up to par? |
| C. Louder than talking | a. Nearly every day |
| ☐ d. Very loud – can be heard in adjacent | b. 3-4 times a week |
| rooms | ☐ c. 1-2 times a week |
| 3. How often do you snore? | d. 1-2 times a month |
| a. Nearly every day | e. Never or nearly never |
| b. 3-4 times a week | 9 Have you ever nedded off or fellen celeen while |
| c. 1-2 times a week | 8. Have you ever nodded off or fallen asleep while driving a vehicle? |
| d. 1-2 times a month | ☐ a. Yes |
| e. Never or nearly never | □ b. No |
| 4. Has your snoring ever bothered other people? | If yes: |
| a. Yes | 9. How often does this occur? |
| □ b. No | |
| C. Don't Know | <ul><li>□ a. Nearly every day</li><li>□ b. 3-4 times a week</li></ul> |
| 5. Has anyone noticed that you quit breathing | c. 1-2 times a week |
| 5. Has anyone noticed that you quit breathing during your sleep? | d. 1-2 times a week |
| a. Nearly every day | e. Never or nearly never |
| b. 3-4 times a week | e. Nevel of hearty nevel |
| c. 1-2 times a week | <u>CATEGORY 3</u> |
| d. 1-2 times a month | 10. Do you have high blood pressure? |
| e. Never or nearly never | Yes |
| <u>-</u> | |
| | ☐ Don't know |
| | _ Zon vallon |

Patient Initials/Signature: \_\_\_\_\_ Date: \_\_\_\_\_

### **BERLIN QUESTIONNAIRE** Height (m) \_\_\_\_\_ Male / Female Weight (kg)\_\_\_\_\_ Age\_\_\_\_ Please choose the correct response to each question. **CATEGORY 1** CATEGORY 2 1. Do you snore? 6. How often do you feel tired or fatigued □ a. Yes after your sleep? □ a. Nearly every day □ b. No □ c. Don't know $\square$ b. 3-4 times a week $\square$ c. 1-2 times a week *If you snore:* $\square$ d. 1-2 times a month □ e. Never or nearly never 2. Your snoring is: □ a. Slightly louder than breathing 7. During your waking time, do you feel tired, fatigued or not up to par? □ b. As loud as talking □ c. Louder than talking □ a. Nearly every day $\Box$ d. Very loud – can be heard in adjacent □ b. 3-4 times a week rooms $\square$ c. 1-2 times a week $\square$ d. 1-2 times a month 3. How often do you snore □ e. Never or nearly never □ a. Nearly every day $\square$ b. 3-4 times a week 8. Have you ever nodded off or fallen asleep while driving a vehicle? $\square$ c. 1-2 times a week □ d. 1-2 times a month □ a. Yes □ b. No □ e. Never or nearly never 4. Has your snoring ever bothered other If yes: people? □ a. Yes 9. How often does this occur? □ b. No □ a. Nearly every day □ c. Don't Know $\square$ b. 3-4 times a week □ c. 1-2 times a week 5. Has anyone noticed that you quit $\square$ d. 1-2 times a month breathing during your sleep? □ e. Never or nearly never

□ a. Nearly every day□ b. 3-4 times a week□ c. 1-2 times a week

□ d. 1-2 times a month□ e. Never or nearly never

### **CATEGORY 3**

| 10. <b>I</b> | Oo you have high blood pressure? |
|--------------|----------------------------------|
| | Yes |
| | No |
| | Don't know |

# Are you Planning to Start Radiation Treatment for Breast Cancer? Worried about Fatigue?

The Dana-Farber Cancer Institute and Brigham and Women's Hospital are seeking *anyone 18 and over beginning radiation treatment for breast cancer* to participate in an observational research study to monitor the development of fatigue during radiation.

Participation includes completion of weekly questionnaires from the start of radiation treatment to 4 weeks after treatment.

If you develop significant fatigue you **may** be eligible for supplemental treatment with an investigational drug.

If you are interested please contact study team at <a href="mailto:DFCIRadiationFatigueStudy@partners.org">DFCIRadiationFatigueStudy@partners.org</a>







# Are you Planning to Start Radiation Treatment for Breast Cancer? Worried about Fatigue?

The Massachusetts General Hospital Cancer Center is seeking *anyone*18 and over beginning radiation treatment for breast cancer to participate in an observational research study to monitor the development of fatigue during radiation.

Participation includes completion of weekly questionnaires from the start of radiation treatment to 4 weeks after treatment.

If you develop significant fatigue you **may** be eligible for supplemental treatment with an investigational drug.

If you are interested please contact:

Lily at 617-726-1923 or email <a href="mailto:ldavis22@partners.org">ldavis22@partners.org</a>
Julia at 617-726-3196 or email <a href="mailto:jdalleva@partners.org">jdalleva@partners.org</a>





| Subject | ID: | | |
|----------|-------|---|---|
| Visit #: | Date: | 1 | 1 |

### **Clinical Variables**

| Radiotherapy-related variables | (to be completed by dosimetrist or physicist): |
|---|---|
| ** | * * * |

| Boost fraction dose (Gy/cGy): Number of boost fractions: Boost target volume (cc): V20, V5 ipsilateral lung (%): | |
|---|---|
| V5 heart (%): | |
| Mean heart dose (cGy): (optional) Volume of tissue receiving 6000 cGy (cc): (optional Volume of tissue receiving 5000 cGy (cc): (optional Volume of tissue receiving 4000 cGy (cc): (optional Volume of tissue receiving 2000 cGy (cc): (optional Volume of tissue receiving 1000 cGy (cc): (optional Volume of tissue receiving 1000 cGy (cc): (optional | )<br><br>) |
| Did subject miss >= 5 scheduled fractions? : yes If yes, Reasons: severe skin reaction Other causes: | ı (yes/No) |
| Did subject miss >= 5 scheduled fractions? : yes | no |
| <u>Dermatologic variables</u> | |
| Fitzpatrick Scale (phototyping): (to be rated by CR | C): |
| type I: white skin, freckles, always burns, never type II: white skin, usually burns, tans minimally type III: cream-white skin, tans uniformly, occas type IV Mediterranean type skin color, rarely burns type V: brown skin, very rarely burns, tans very type VI: very dark brown to black skin, never bu | ionally burns<br>rns, always tans well<br>easily |

| | | | | Subject ID | : | | |
|---|---|---|---|---|---|---|---|
| | | | | Subject ID<br>Visit #: | Date: | _/ | / |
| De | mographic Information | | | | | | |
| Αg | e: Date of Birth:/ | _/_ | | | | | |
| Wi | th what racial groups do you most closely identify? | | | | | | |
| | White/Caucasian | | | | | | |
| | Black or African-American | | | | | | |
| | Asian | | | | | | |
| | Native Hawaiian or other Pacific Islander | | | | | | |
| | Other (please specify) | | | | | | |
| | American Indian or Alaska Native | | | | | | |
| | Decline to answer | | | | | | |
| Wi | th what ethnic groups do you most closely identify? | | | | | | |
| | Hispanic/Latina | | | | | | |
| | Non-Hispanic/ Non-Latina | | | | | | |
| | Decline to answer | | | | | | |
| | Decime to diamet | | | | | | |
| W | nat is your marital status? | | | | | | |
| | Single (Never married) | | | | | | |
| | Divorced/ Separated | | | | | | |
| | Married | | | | | | |
| | Widowed | | | | | | |
| | Living in a marriage-like relationship | | | | | | |
| W | nat is the highest level of schooling you have complet | ed? | | | | | |
| | Didn't go to high school | | | | | | |
| | Some high school | | | | | | |
| | High school diploma or GED | | | | | | |
| | Some college or technical school | | | | | | |
| | Graduated college (4 year college degree) | | | | | | |
| | Complete Graduate School | | | | | | |
| En | ployment Status (check all that apply) | | | | | | |
| | Full-time | П | Homemaker | | | | |
| | Student | | Disabled | | | | |
| | Part-time | | Unemployed | | | | |
| | Retired | | Other, please sp | recify. | | | |
| | Retified | ш | omer, piease sp | CC11y | | | |
| Нс | w many live births have you had? | _ | | | | | |

| How many children do you have living at home? |
|---|
| Cigarette smoking: |
| □ Never |
| ☐ Former, quit date ☐ ☐ / ☐ ☐ ☐ (month, year) |
| ☐ Current (# Cigarettes/ day) |
| Current alcohol consumption: |
| □ No |
| ☐ Yes (Drinks/week) |
| What is your travel time to the radiation clinic (in minutes)? |
| How much do you exercise, in a manner that raises your heart rate (average number of minutes per week)? |
| How much exposure to the sun have you gotten over the last month (average number of minutes per day)? |
| Do you wear sunscreen and/or protective clothing when exposed to sun? |
| What is your natural hair color? |
| Menopause |
| When was your last menstrual period? |
| Month Year |
| Have you had a menstrual period in the last 5 months? |
| □ No |
| □ Yes |
| Did your menses stop or become irregular during chemotherapy? |
| □ No |
| □ Yes |
| □ Not applicable |

Subject ID: \_\_\_\_\_ Visit #:\_\_\_\_ Date: \_\_\_\_/\_

| | | Subject IE | ):<br>Date: | | |
|---|---|---|---|---|---|
| | | Visit #: | _ Date: | / | _′ |
| Но | w old were you when you first started having hot flashes? | | | | |
| | Never had hot flashes | | | | |
| | years old | | | | |
| | what point did you begin having hot flashes? (Check all that apply.) Never had hot flashes When menstrual periods became irregular Had a hysterectomy When both ovaries were removed During or after chemotherapy After anti-estrogen therapy (Tamoxifen, Evista, Femara, Arimidex, Arom Don't know Other (specify) | nasin) was | started | | |
| Ha<br>□ | tigue ve you ever had fatigue BEFORE breast cancer that interfered with No Yes | your daily | activities | ;? | |
| Ple | ves -> ves answer the following questions related to the period of MOST SEVER the past. | E fatigue y | ou experie | enced | |
| Но | w old were you when you had this fatigue? | | | | |
| Но | w long did it last? (in months) | | | | |
| If y | yes, what was the cause of the fatigue (check any/all that apply)?: Insomnia or sleep apnea | | | | |
| | Thyroid problems | | | | |
| | Menopause | | | | |
| | Stress or anxiety | | | | |
| | Depression | | | | |
| | Infection | | | | |
| | Asthma or allergies | | | | |
| | Anemia | | | | |
| | Don't know | | | | |
| | Other (specify) | | | | |

| | Subject II | D: | |
|---|---|---|---|
| | Visit#: | D:<br>Date: | / |
| Other medical problems | | | |
| Have you ever experienced any of the following conditions: | | | |
| ☐ Insomnia | | | |
| ☐ Sleep apnea | | | |
| ☐ Thyroid problems | | | |
| □ Diabetes | | | |
| ☐ High blood pressure | | | |
| ☐ Depression | | | |
| ☐ Anxiety | | | |
| ☐ Anemia | | | |
| ☐ Asthma or allergies | | | |
| ☐ Other medical condition (specify) | | | |
| Depression | | | |
| Has a medical professional or mental health provider ever told you that yo | ou had depress | sion? | |
| □ No | | | |
| Yes | : 1 4 . 1 | | |
| How old were you when you first saw a doctor or other clinic years old | ian about dep | ression? | |
| How old were you when you last saw a doctor or other clinici years old | an about depi | ession? | |
| Was your depression diagnosed BEFORE your breast cancer? □ No □ Yes | | | |
| Have you ever been treated for depression? | | | |
| □ No | | | |
| ☐ Yes | | | |
| If yes, what were you treated with? | | | |
| ☐ Antidepressant | | | |
| ☐ Therapy | | | |
| Other (specify) | | | |
| Patient Initials/Signature: | | | |
| | Date: | · | |

Naltrexone RCT for Treatment-Emergent Fatigue in Women Receiving Radiation Therapy for Breast Cancer Protocol 14-056 PI: Fremonta Meyer MD Subject Exit Form Subject ID: \_\_\_\_ Date: / / Date of study termination (or last correspondence, if lost to follow-up): \_\_\_/ \_\_\_/ Last Visit Completed: \_\_\_\_ **Did subject receive study drug?** Yes No Was the subject eligible for the intervention phase? ☐yes ☐no Reason for ineligibility: FACIT-F drop of less than 10 points during radiotherapy FACIT –F <=10 prior to radiotherapy Major depression and/or suicidal ideation on PHQ9 (please circle which) Recent use of opioids or expected requirement for opioids Abnormal lab values (please specify which:) Other: (please specify) If ineligible for the intervention, did the subject complete the entire monitoring phase? ves no Reason for exiting either phase of study:

Reason for exiting either phase of study:

\_\_\_\_ Requirement for opioids \_\_\_\_ Geographic relocation

\_\_\_ Lost to follow up \_\_\_\_ Development of medical safety issues

\_\_\_ Loss of interest \_\_\_\_ Noncompliance with visits

\_\_\_ Too much time involved for participation

Other (please specify): Adverse event

Comment on reason for exiting study (optional):\_\_\_\_\_

| Nattrexone RC1 for Treatment-Emergent | t Fatigue in Women Receiving Radiation Therapy for Breast |
|---|---|
| Cancer | |
| Protocol 14-056 | |
| PI: Fremonta Meyer MD Who initiated termination: Clin | nician Subject |
| Form completed by: | Date:/ |
| DA/DI Signaturo: | Date: / / |

| Patient ID: |
|-------------|
| Date: |
| Visit#: |

### **FACIT Fatigue Scale (Version 4)**

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the <u>past 7 days</u>.

| | | Not at | A<br>little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| 1 | I feel fatigued | 0 | 1 | 2 | 3 | 4 |
| 2 | I feel weak all over | 0 | 1 | 2 | 3 | 4 |
| 3 | I feel listless ("washed out") | 0 | 1 | 2 | 3 | 4 |
| 4 | I feel tired | 0 | 1 | 2 | 3 | 4 |
| 5 | I have trouble starting things because I am tired | 0 | 1 | 2 | 3 | 4 |
| 6 | I have trouble finishing things because I am tired | 0 | 1 | 2 | 3 | 4 |
| 7 | I have energy | 0 | 1 | 2 | 3 | 4 |
| 8 | I am able to do my usual activities | 0 | 1 | 2 | 3 | 4 |
| 9 | I need to sleep during the day | 0 | 1 | 2 | 3 | 4 |
| 10 | I am too tired to eat | 0 | 1 | 2 | 3 | 4 |
| 11 | I need help doing my usual activities | 0 | 1 | 2 | 3 | 4 |
| 12 | I am frustrated by being too tired to do the things I want to do | 0 | 1 | 2 | 3 | 4 |
| 13 | I have to limit my social activity because I am tired | 0 | 1 | 2 | 3 | 4 |

| Patient Initials/Signature: |
|-----------------------------|
| Date: |